CLINICAL TRIAL: NCT05827926
Title: A Phase 1/2, Randomized, Observer-blind, Active-Control Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-based Influenza and SARS-CoV-2 Multi-component Vaccines in Healthy Adults
Brief Title: A Study of mRNA-based Influenza and SARS-CoV-2 (COVID-19) Multi-component Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1083-P101
Record Dates: First submitted 2023-04-24; First posted 2023-04-25 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2; Influenza
Keywords: mRNA-1083; mRNA-1083 Vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; Influenza Vaccine; Moderna; Influenza
MeSH Terms: conditions — Influenza, Human; Coronavirus Infections; Virus Diseases | interventions — Baiya SARS-CoV-2 VAX COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (37):
- Part 1 Cohort A2: mRNA-1083.1 Dose B (Experimental): Participants will receive single intramuscular (IM) injection of mRNA-1083.1 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083.1
- Part 1 Cohort A3: mRNA-1083.1 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083.1 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083.1
- Part 1 Cohort A4: mRNA-1083.2 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort A5: mRNA-1083.2 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort A6: mRNA-1083.2 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort A7: mRNA-1083.3 (Experimental): Participants will receive single IM injection of mRNA-1083.3 on Day 1.
  Interventions: Biological: mRNA-1083.3
- Part 1 Cohort A8: Investigational Influenza Vaccine 1 (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 1 on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 1
- Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 (Active Comparator): Participants will receive single IM injection of Investigational COVID-19 Vaccine 1 on Day 1.
  Interventions: Biological: Investigational COVID-19 Vaccine 1
- Part 1 Cohort A10: COVID-19 Vaccine 1 (Active Comparator): Participants will receive single IM injection of COVID-19 Vaccine 1 on Day 1.
  Interventions: Biological: COVID-19 Vaccine 1
- Part 1 Cohort A11: Investigational Influenza Vaccine 2 (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 2 on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 2
- Part 1 Cohort A12: Influenza Vaccine 1 (Active Comparator): Participants will receive single IM injection of Influenza Vaccine 1 on Day 1.
  Interventions: Biological: Influenza Vaccine 1
- Part 1 Cohort A13: Influenza Vaccine 2 (Active Comparator): Participants will receive single IM injection of Influenza Vaccine 2 on Day 1.
  Interventions: Biological: Influenza Vaccine 2
- Part 1 Cohort B1: mRNA-1083.1 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083.1 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083.1
- Part 1 Cohort B2: mRNA-1083.1 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083.1 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083.1
- Part 1 Cohort B3: mRNA-1083.1 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083.1 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083.1
- Part 1 Cohort B4: mRNA-1083.2 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort B5: mRNA-1083.2 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort B6: mRNA-1083.2 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083.2 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083.2
- Part 1 Cohort B7: mRNA-1083.3 (Experimental): Participants will receive single IM injection of mRNA-1083.3 on Day 1.
  Interventions: Biological: mRNA-1083.3
- Part 1 Cohort B8: Investigational Influenza Vaccine 1 (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 1 on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 1
- Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 (Active Comparator): Participants will receive single IM injection of Investigational COVID-19 Vaccine 1 on Day 1.
  Interventions: Biological: Investigational COVID-19 Vaccine 1
- Part 1 Cohort B10: COVID-19 Vaccine 1 (Active Comparator): Participants will receive single IM injection of COVID-19 Vaccine 1 on Day 1.
  Interventions: Biological: COVID-19 Vaccine 1
- Part 1 Cohort B11: Investigational Influenza Vaccine 2 (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 2 on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 2
- Part 1 Cohort B12: Influenza Vaccine 1 (Active Comparator): Participants will receive single IM injection of Influenza Vaccine 1 on Day 1.
  Interventions: Biological: Influenza Vaccine 1
- Part 2: mRNA-1083 Composition 1 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 2 Dose A (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level A on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 1 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 2 Dose B (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level B on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 1 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 2 Dose C (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level C on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 1 Dose D (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 1 at Dose Level D on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: mRNA-1083 Composition 2 Dose D (Experimental): Participants will receive single IM injection of mRNA-1083 Composition 2 at Dose Level D on Day 1.
  Interventions: Biological: mRNA-1083
- Part 2: Investigational Influenza Vaccine 1 Dose A (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 1 at Dose Level A on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 1
- Part 2: Investigational Influenza Vaccine 1 Dose B (Active Comparator): Participants will receive single IM injection of Investigational Influenza Vaccine 1 at Dose Level B on Day 1.
  Interventions: Biological: Investigational Influenza Vaccine 1
- Part 2: Investigational COVID-19 Vaccine 2 (Active Comparator): Participants will receive single IM injection of Investigational COVID-19 Vaccine 2 on Day 1.
  Interventions: Biological: Investigational COVID-19 Vaccine 2
- Part 2: COVID-19 Vaccine 2 (Active Comparator): Participants will receive single IM injection of COVID-19 Vaccine 2 on Day 1.
  Interventions: Biological: COVID-19 Vaccine 2
- Part 2: Influenza Vaccine 1 (Active Comparator): Participants will receive single IM injection of Influenza Vaccine 1 on Day 1.
  Interventions: Biological: Influenza Vaccine 1

INTERVENTIONS:
Biological: Influenza Vaccine 1 — quadrivalent seasonal influenza vaccine
  Arms: Part 1 Cohort A12: Influenza Vaccine 1; Part 1 Cohort B12: Influenza Vaccine 1; Part 2: Influenza Vaccine 1
Biological: mRNA-1083.1 — Sterile liquid for injection
  Arms: Part 1 Cohort A2: mRNA-1083.1 Dose B; Part 1 Cohort A3: mRNA-1083.1 Dose C; Part 1 Cohort B1: mRNA-1083.1 Dose A; Part 1 Cohort B2: mRNA-1083.1 Dose B; Part 1 Cohort B3: mRNA-1083.1 Dose C
Biological: mRNA-1083.2 — Sterile liquid for injection
  Arms: Part 1 Cohort A4: mRNA-1083.2 Dose A; Part 1 Cohort A5: mRNA-1083.2 Dose B; Part 1 Cohort A6: mRNA-1083.2 Dose C; Part 1 Cohort B4: mRNA-1083.2 Dose A; Part 1 Cohort B5: mRNA-1083.2 Dose B; Part 1 Cohort B6: mRNA-1083.2 Dose C
Biological: mRNA-1083.3 — Sterile liquid for injection
  Arms: Part 1 Cohort A7: mRNA-1083.3; Part 1 Cohort B7: mRNA-1083.3
Biological: Investigational Influenza Vaccine 1 — Sterile liquid for injection
  Arms: Part 1 Cohort A8: Investigational Influenza Vaccine 1; Part 1 Cohort B8: Investigational Influenza Vaccine 1; Part 2: Investigational Influenza Vaccine 1 Dose A; Part 2: Investigational Influenza Vaccine 1 Dose B
Biological: Investigational COVID-19 Vaccine 1 — Sterile liquid for injection
  Arms: Part 1 Cohort A9: Investigational COVID-19 Vaccine 1; Part 1 Cohort B9: Investigational COVID-19 Vaccine 1
Biological: COVID-19 Vaccine 1 — Sterile liquid for injection
  Arms: Part 1 Cohort A10: COVID-19 Vaccine 1; Part 1 Cohort B10: COVID-19 Vaccine 1
Biological: Investigational Influenza Vaccine 2 — Sterile liquid for injection
  Arms: Part 1 Cohort A11: Investigational Influenza Vaccine 2; Part 1 Cohort B11: Investigational Influenza Vaccine 2
Biological: Influenza Vaccine 2 — quadrivalent seasonal influenza vaccine
  Arms: Part 1 Cohort A13: Influenza Vaccine 2
Biological: mRNA-1083 — Sterile liquid for injection
  Arms: Part 2: mRNA-1083 Composition 1 Dose A; Part 2: mRNA-1083 Composition 1 Dose B; Part 2: mRNA-1083 Composition 1 Dose C; Part 2: mRNA-1083 Composition 1 Dose D; Part 2: mRNA-1083 Composition 2 Dose A; Part 2: mRNA-1083 Composition 2 Dose B; Part 2: mRNA-1083 Composition 2 Dose C; Part 2: mRNA-1083 Composition 2 Dose D
Biological: Investigational COVID-19 Vaccine 2 — Sterile liquid for injection
  Arms: Part 2: Investigational COVID-19 Vaccine 2
Biological: COVID-19 Vaccine 2 — Sterile liquid for injection
  Arms: Part 2: COVID-19 Vaccine 2

SUMMARY:
The study is divided into 2 parts: Part 1 and Part 2. The purpose of Part 1 of this study is to generate sufficient safety, reactogenicity, and immunogenicity data to enable selection of an mRNA-1083 vaccine composition and dose level to evaluate in a subsequent Phase 3 clinical trial in adults.

The purpose of Part 2 of this study is to generate safety and immunogenicity data for additional mRNA-1083 compositions and dose levels in young adults ≥18 years and <50 years of age.

DETAILED DESCRIPTION:
Part 1: Participants will be enrolled into 1 of 2 age cohorts: Cohort A for adults ≥65 to <80 years of age or Cohort B for adults ≥18 to <65 year of age. In Cohort A, approximately 600 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since September 2022). In Cohort B, approximately 624 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by 2 age groups: ≥18 to <50 years and ≥50 to <65 years of age and by influenza vaccine status in the most recent influenza season (received or not received since September 2022).

Part 2: Approximately, 520 participants between ≥18 to <50 years of age will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since Sept 2023).

ELIGIBILITY:
Key Inclusion Criteria:

Part 1 (Phase 1/2)

* Adults ≥18 to <80 years of age at the time of consent.
* Body mass index (BMI) of 18 kilograms (kg)/square meter (m^2) to 35 kg/m^2 (inclusive) at the Screening Visit.
* Healthy as determined by medical evaluation, including medical history, physical examination, and laboratory tests.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 90 days following vaccine administration, and not currently breastfeeding.
* Fully vaccinated for COVID-19 primary series according to the locally authorized or approved regimen, and their last COVID-19 vaccine (primary series or booster) was ≥120 days prior to Day 1.

Part 2 (Phase 2 Extension)

* Adults ≥18 to <50 years of age at the time of consent.
* BMI of 18 kg/m^2 to 35 kg/m^2 (inclusive) at the Screening Visit.
* Healthy as determined by medical evaluation, including medical history, and physical examination.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 90 days following vaccine administration, and not currently breastfeeding.
* Have received at least 2 doses of locally authorized or approved COVID-19 vaccines and last dose was ≥90 days prior to Day 1.

Key Exclusion Criteria:

Part 1 (Phase 1/2) and Part 2 (Phase 2 Extension)

* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the clinical trial or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants for >14 days in total within 180 days prior to Screening Visit (for glucocorticoids ≥10 milligrams [mg]/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the clinical trial (including intra-articular steroid injections). Inhaled, nasal, and topical steroids are allowed.
* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to study intervention administration or plans to receive a vaccine authorized or approved by a local health agency within 28 days after study intervention administration.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine within 150 days prior to Day 1.
* Participant tested positive for influenza by local health authority-approved testing methods ≤150 days prior to Day 1.
* Participant has had close contact to someone with COVID-19 as defined by the Centers for Disease Control and Prevention (CDC) in the past 10 days prior to Day 1.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the clinical trial.
* Working or has worked as study personnel, is an immediate family member or household member of study personnel, study site staff, or Sponsor personnel, or resides in a nursing home.

Part 2 (Phase 2 Extension) Only

* Participants who enrolled in Part 1 of the mRNA-1083-P101 (Phase 1/2) study.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1758 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Chandler Clinical Trials, Chandler, Arizona
  - Benchmark Research, Colton, California
  - Marvel Clinical Research, Huntington Beach, California
  - Central Valley Research, Modesto, California
  - Benchmark Research, Sacramento, California
  - Tekton Research, Longmont, Colorado
  - Accel Research Sites, DeLand, Florida
  - CenExel, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Accel Research Sites, Maitland, Florida
  - Suncoast Research Group, Miami, Florida
  - Centricity Research, Columbus, Georgia
  - Accel Research Site, Decatur, Georgia
  - CenExel iResearch, Decatur, Georgia
  - Lifeline Primary Care, Lilburn, Georgia
  - Koch Family Medicine, Morton, Illinois
  - Optimal Research, Peoria, Illinois
  - DM Clinical Research, River Forest, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Tekton Research, Wichita, Kansas
  - Versailles Family Medicine, Versailles, Kentucky
  - Velocity Clinical research, Baton Rouge, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Annapolis Internal Medicine, Annapolis, Maryland
  - Velocity Clinical Research, Rockville, Maryland
  - DM Clinical Research, Brookline, Massachusetts
  - Vida Clinical Studies, Dearborn Heights, Michigan
  - DelRicht Research, Gulfport, Mississippi
  - Clay Platte Family Medicine, Kansas City, Missouri
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - CCT Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - Tryon Medical Partners, Charlotte, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Centricity Research, Columbus, Ohio
  - WellNow Urgent Care & Research, Dayton, Ohio
  - Lynn Institute of East Oklahoma, Oklahoma City, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Tekton Research Inc, Yukon, Oklahoma
  - DM Clinical Research, Philadelphia, Pennsylvania
  - Mercado Medical Practice, Philadelphia, Pennsylvania
  - DelRicht Research, Charleston, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Medical Care, Elizabethton, Tennessee
  - DelRicht Research, Hendersonville, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Tekton Research, Beaumont, Texas
  - Benchmark Research, Fort Worth, Texas
  - Cyfair Clinical Research, Houston, Texas
  - Texas Center for Drug Development, Houston, Texas
  - DelRicht Research, McKinney, Texas
  - Benchmark Research, San Angelo, Texas
  - Tekton Research, San Antonio, Texas
  - CCT Research, Pleasant View, Utah
  - Ogden Clinic, Roy, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - Meridian Clinical Research, Hampton, Virginia
  - Velocity Clinical Research, Portsmouth, Virginia
  - Wenatchee Valley Hospital & Clinics Campus, Wenatchee, Washington

REFERENCES:
- [Derived] Rudman Spergel AK, Ananworanich J, Guo R, Deng W, Carmona L, Schaefers K, Paila YD, Kandinov B, Eger CH, Sinkiewicz M, Shao S, Henry C, Shaw CA. mRNA-based seasonal influenza and SARS-CoV-2 multicomponent vaccine in healthy adults: a phase 1/2 trial. Nat Med. 2025 May;31(5):1484-1493. doi: 10.1038/s41591-025-03591-0. Epub 2025 Mar 18. PMID 40102593

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Cohort A12: Influenza Vaccine 1; Part 1 Cohort B12: Influenza Vaccine 1; Part 2: Influenza Vaccine 1: Participants received a single IM injection of Influenza Vaccine 1 on Day 1.
- Part 1 Cohort A13: Influenza Vaccine 2: Participants received a single IM injection of Influenza Vaccine 2 on Day 1.
- Part 1 Cohort A11: Investigational Influenza Vaccine 2; Part 1 Cohort B11: Investigational Influenza Vaccine 2: Participants received a single IM injection of Investigational Influenza Vaccine 2 on Day 1.
- Part 1 Cohort A8: Investigational Influenza Vaccine 1; Part 1 Cohort B8: Investigational Influenza Vaccine 1: Participants received a single IM injection of Investigational Influenza Vaccine 1 on Day 1.
- Part 1 Cohort A10: COVID-19 Vaccine 1; Part 1 Cohort B10: COVID-19 Vaccine 1: Participants received a single IM injection of COVID-19 Vaccine 1 on Day 1.
- Part 1 Cohort A9: Investigational COVID-19 Vaccine 1; Part 1 Cohort B9: Investigational COVID-19 Vaccine 1: Participants received a single IM injection of Investigational COVID-19 Vaccine 1 on Day 1.
- Part 1 Cohort A2: mRNA-1083.1 Dose Level 2; Part 1 Cohort B2: mRNA-1083.1 Dose Level 2: Participants received a single IM injection of mRNA-1083.1 at dose level 2 on Day 1.
- Part 1 Cohort A3: mRNA-1083.1 Dose Level 3; Part 1 Cohort B3: mRNA-1083.1 Dose Level 3: Participants received a single IM injection of mRNA-1083.1 at dose level 3 on Day 1.
- Part 1 Cohort A4: mRNA-1083.2 Dose Level 1; Part 1 Cohort B4: mRNA-1083.2 Dose Level 1: Participants received a single IM injection of mRNA-1083.2 at dose level 1 on Day 1.
- Part 1 Cohort A5: mRNA-1083.2 Dose Level 2; Part 1 Cohort B5: mRNA-1083.2 Dose Level 2: Participants received a single IM injection of mRNA-1083.2 at dose level 2 on Day 1.
- Part 1 Cohort A6: mRNA-1083.2 Dose Level 3; Part 1 Cohort B6: mRNA-1083.2 Dose Level 3: Participants received a single IM injection of mRNA-1083.2 at dose level 3 on Day 1.
- Part 1 Cohort A7: mRNA-1083.3; Part 1 Cohort B7: mRNA-1083.3: Participants received a single IM injection of mRNA-1083.3 on Day 1.
- Part 1 Cohort B1: mRNA-1083.1 Dose Level 1: Participants received a single IM injection of mRNA-1083.1 at dose level 1 on Day 1.
- Part 2: Investigational Influenza Vaccine 1 Dose Level 1: Participants received a single IM injection of Investigational Influenza Vaccine 1 at dose level 1 on Day 1.
- Part 2: Investigational Influenza Vaccine 1 Dose Level 2: Participants received a single IM injection of Investigational Influenza Vaccine 1 at dose level 2 on Day 1.
- Part 2: COVID-19 Vaccine 2: Participants received a single IM injection of COVID-19 Vaccine 2 on Day 1.
- Part 2: Investigational COVID-19 Vaccine 2: Participants received a single IM injection of Investigational COVID-19 Vaccine 2 on Day 1.
- Part 2: mRNA-1083 Composition 1 Dose Level 1: Participants received a single IM injection of mRNA-1083 Composition 1 at dose level 1 on Day 1.
- Part 2: mRNA-1083 Composition 1 Dose Level 2: Participants received a single IM injection of mRNA-1083 Composition 1 at dose level 2 on Day 1.
- Part 2: mRNA-1083 Composition 1 Dose Level 3: Participants received a single IM injection of mRNA-1083 Composition 1 at dose level 3 on Day 1.
- Part 2: mRNA-1083 Composition 1 Dose Level 4: Participants received a single IM injection of mRNA-1083 Composition 1 at dose level 4 on Day 1.
- Part 2: mRNA-1083 Composition 2 Dose Level 1: Participants received a single IM injection of mRNA-1083 Composition 2 at dose level 1 on Day 1.
- Part 2: mRNA-1083 Composition 2 Dose Level 2: Participants received a single IM injection of mRNA-1083 Composition 2 at dose level 2 on Day 1.
- Part 2: mRNA-1083 Composition 2 Dose Level 3: Participants received a single IM injection of mRNA-1083 Composition 2 at dose level 3 on Day 1.
- Part 2: mRNA-1083 Composition 2 Dose Level 4: Participants received a single IM injection of mRNA-1083 Composition 2 at dose level 4 on Day 1.
Period: Overall Study
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Started | 54 | 53 | 54 | 53 | 54 | 52 | 52 | 33 | 54 | 54 | 33 | 53 | 52 | 56 | 56 | 56 | 55 | 56 | 56 | 37 | 55 | 56 | 38 | 56 | 41 | 40 | 40 | 42 | 40 | 40 | 42 | 42 | 41 | 40 | 40 | 40 | 42
Received Study Injection | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 54 | 54 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 55 | 56 | 37 | 55 | 55 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Safety Set (All randomized participants who received the study intervention. Participants were included in the vaccination group corresponding to what they actually received (as treated).) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 55 | 53 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 56 | 55 | 37 | 56 | 54 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Solicited Safety Set (All randomized participants who received the study intervention and contributed any solicited adverse reaction (AR) data. Participants were included in the vaccination group corresponding to what they actually received (as treated).) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 55 | 53 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 56 | 55 | 37 | 56 | 54 | 38 | 53 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Per Protocol Set (All randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response. Participants were analyzed according to group to which they were randomized.) | 51 | 50 | 50 | 45 | 51 | 49 | 50 | 30 | 53 | 51 | 31 | 50 | 50 | 48 | 52 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 51 | 38 | 38 | 37 | 40 | 38 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
Full Analysis Set (FAS) (All randomized participants who received the study intervention. Participants were analyzed according to the group to which they were randomized.) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 54 | 54 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 55 | 56 | 37 | 55 | 55 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Completed | 52 | 53 | 53 | 51 | 54 | 51 | 51 | 33 | 54 | 54 | 33 | 53 | 50 | 53 | 55 | 52 | 52 | 55 | 55 | 37 | 53 | 53 | 36 | 53 | 38 | 38 | 36 | 40 | 38 | 39 | 37 | 39 | 38 | 38 | 39 | 37 | 37
Not Completed | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 4 | 3 | 1 | 1 | 0 | 2 | 3 | 2 | 3 | 3 | 2 | 4 | 2 | 2 | 1 | 5 | 3 | 3 | 2 | 1 | 3 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 4 | 1 | 2 | 1 | 5 | 0 | 3 | 2 | 1 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Other Than Specified | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The FAS included all randomized participants who received the study intervention. Participants were analyzed according to the group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4 | Total
Number analyzed (Participants) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 54 | 54 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 55 | 56 | 37 | 55 | 55 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42 | 1743
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 52 | 55 | 55 | 53 | 55 | 55 | 56 | 37 | 55 | 55 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42 | 1147
  >=65 years | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 54 | 54 | 33 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 596
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 29 | 29 | 33 | 30 | 27 | 16 | 30 | 30 | 14 | 28 | 32 | 23 | 31 | 29 | 28 | 28 | 31 | 17 | 33 | 31 | 24 | 30 | 23 | 20 | 24 | 18 | 15 | 22 | 21 | 22 | 18 | 23 | 25 | 22 | 23 | 941
  Male | 22 | 23 | 25 | 22 | 21 | 22 | 24 | 17 | 24 | 24 | 19 | 25 | 20 | 32 | 24 | 24 | 27 | 27 | 25 | 20 | 22 | 24 | 14 | 24 | 17 | 19 | 16 | 24 | 25 | 18 | 21 | 19 | 23 | 17 | 15 | 18 | 19 | 802
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 6 | 3 | 4 | 6 | 8 | 4 | 5 | 4 | 3 | 8 | 8 | 2 | 8 | 7 | 4 | 7 | 5 | 5 | 9 | 7 | 5 | 5 | 7 | 3 | 4 | 2 | 8 | 4 | 10 | 11 | 2 | 5 | 10 | 6 | 6 | 209
  Not Hispanic or Latino | 50 | 49 | 47 | 47 | 50 | 44 | 43 | 28 | 49 | 49 | 30 | 45 | 44 | 51 | 47 | 46 | 51 | 47 | 50 | 32 | 46 | 48 | 33 | 48 | 33 | 35 | 36 | 40 | 32 | 35 | 32 | 29 | 38 | 34 | 30 | 34 | 35 | 1517
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 48 | 47 | 46 | 44 | 44 | 43 | 46 | 28 | 45 | 50 | 27 | 45 | 38 | 39 | 43 | 36 | 37 | 36 | 37 | 30 | 41 | 39 | 22 | 37 | 29 | 26 | 25 | 26 | 25 | 29 | 26 | 24 | 24 | 22 | 22 | 22 | 29 | 1277
  Race: Black or African American | 6 | 5 | 8 | 6 | 9 | 7 | 5 | 5 | 5 | 4 | 6 | 6 | 13 | 12 | 7 | 14 | 12 | 11 | 16 | 3 | 11 | 11 | 14 | 14 | 7 | 7 | 12 | 10 | 7 | 6 | 10 | 10 | 9 | 13 | 7 | 13 | 9 | 330
  Race: Asian | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 3 | 4 | 2 | 3 | 0 | 4 | 1 | 2 | 4 | 6 | 3 | 5 | 4 | 3 | 4 | 5 | 6 | 3 | 7 | 3 | 3 | 90
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Race: Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 14
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 14
  Race: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race: Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were reported by participants an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills.
Time Frame: Up to 7 days after study injection
Population: The solicited safety set included all randomized participants who receive the study intervention and contribute any solicited AR data. Participants were included in the vaccination group corresponding to what they actually received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 55 | 53 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 56 | 55 | 37 | 56 | 54 | 38 | 53 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Participants | 32 | 36 | 37 | 43 | 42 | 31 | 44 | 26 | 42 | 46 | 29 | 46 | 33 | 49 | 51 | 46 | 41 | 47 | 50 | 34 | 46 | 51 | 38 | 47 | 32 | 32 | 39 | 40 | 34 | 34 | 39 | 37 | 38 | 33 | 34 | 37 | 39

2. Primary Outcome: Parts 1 and 2: Number of Participants With Unsolicited Adverse Events (AEs) and Severe AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Severity for all unsolicited AEs was determined by the Investigator based upon medical judgment and graded as Mild, Moderate or Severe. Number of participants with unsolicited AEs (SAEs and non-serious AEs) and severe AEs up to 28 days post-vaccination are reported in this outcome measure. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 28 days after study injection
Population: The Safety Set included all randomized participants who received the study intervention. Participants were included in the vaccination group corresponding to what they actually received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 55 | 53 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 56 | 55 | 37 | 56 | 54 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Participants
  Unsolicited AEs | 5 | 9 | 7 | 5 | 7 | 9 | 7 | 2 | 6 | 6 | 5 | 8 | 5 | 11 | 8 | 9 | 8 | 11 | 6 | 6 | 6 | 8 | 8 | 5 | 5 | 3 | 6 | 4 | 4 | 4 | 3 | 3 | 6 | 5 | 4 | 5 | 8
  Severe AEs | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Parts 1 and 2: Number of Participants With Unsolicited Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Study Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs were protocol-defined medical concepts. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or COVID-19 and visits to healthcare practitioners external to the study site. Number of participants with SAEs, AESIs, MAAEs, and AEs leading to study discontinuation up to Day 181 are reported in this outcome measure. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 181
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 54 | 53 | 54 | 51 | 54 | 52 | 51 | 33 | 55 | 53 | 33 | 53 | 52 | 55 | 55 | 53 | 55 | 56 | 55 | 37 | 56 | 54 | 38 | 54 | 40 | 39 | 40 | 42 | 40 | 40 | 42 | 41 | 41 | 40 | 40 | 40 | 42
Participants
  SAEs | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  AESIs | 3 | 1 | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  MAAEs | 11 | 16 | 13 | 16 | 13 | 20 | 12 | 4 | 12 | 14 | 7 | 10 | 13 | 13 | 13 | 17 | 17 | 15 | 10 | 9 | 10 | 13 | 12 | 5 | 8 | 7 | 6 | 8 | 8 | 10 | 6 | 11 | 6 | 11 | 10 | 9 | 8
  AEs Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Geometric Mean Titer (GMT) of Antibodies for Influenza at Day 29, as Measured by Hemagglutination Inhibition (HAI) Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5 * LLOQ. Values greater than the upper limit of quantification (ULOQ) were converted to the ULOQ. LLOQ = 10 and ULOQ = 3620 for Influenza A H1N1 antibody, LLOQ = 10 and ULOQ = 5120 for Influenza A H3N2 antibody, LLOQ = 10 and ULOQ = 1356 for Influenza B/Victoria-lineage antibody, and LLOQ = 10 and ULOQ = 1280 for Influenza B/Yamagata-lineage antibody. 95% confidence interval (CI) was calculated based on the t-distribution of the log-transformed values for geometric mean (GM) titer, then back transformed to the original scale for presentation. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Day 29
Population: PP Set included all randomized participants who received the study intervention, complied with the injection schedule, complied with the timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected the immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 38 | 38 | 37 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
titer
  Influenza A H1N1 Antibody | 80.0 [50.3 to 127.2] | 105.1 [71.9 to 153.7] | 129.0 [86.2 to 193.1] | 73.9 [52.6 to 103.6] | 98.3 [71.3 to 135.5] | 111.2 [81.2 to 152.5] | 99.9 [69.6 to 143.4] | 85.7 [61.0 to 120.4] | 88.4 [64.3 to 121.5] | 71.2 [47.6 to 106.7] | 106.0 [73.3 to 153.2]
  Influenza A H3N2 Antibody | 80.7 [60.9 to 107.0] | 96.0 [66.3 to 139.1] | 155.6 [111.4 to 217.3] | 65.8 [50.3 to 86.1] | 71.3 [53.9 to 94.2] | 105.6 [80.2 to 139.0] | 79.3 [59.5 to 105.7] | 62.2 [45.5 to 85.1] | 79.3 [61.8 to 101.7] | 75.2 [54.0 to 104.5] | 80.7 [64.5 to 100.8]
  Influenza B/Victoria-lineage Antibody | 86.0 [67.7 to 109.2] | 80.7 [59.5 to 109.5] | 141.9 [100.3 to 200.8] | 75.8 [57.4 to 100.2] | 104.2 [81.1 to 133.8] | 108.4 [84.2 to 139.5] | 106.3 [76.4 to 147.9] | 98.5 [72.2 to 134.3] | 78.5 [61.3 to 100.6] | 75.9 [56.7 to 101.6] | 82.0 [63.8 to 105.5]
  Influenza B/Yamagata-lineage Antibody | 140.8 [110.2 to 179.9] | 122.8 [99.2 to 151.9] | 179.0 [130.4 to 245.7] | 80.7 [64.1 to 101.7] | 101.6 [80.0 to 129.0] | 112.2 [87.8 to 143.3] | 112.2 [90.1 to 139.7] | 94.3 [69.6 to 127.9] | 118.3 [87.4 to 160.3] | 97.7 [74.8 to 127.5] | 98.3 [76.5 to 126.2]

5. Primary Outcome: Part 2: GM Concentration of Antibodies for SARS-CoV-2 at Day 29, as Measured by Pseudovirus Neutralization Assay (PsVNA)
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Antibody values reported as below the LLOQ are replaced by 0.5 * LLOQ. Values greater than the ULOQ are converted to the ULOQ. LLOQ = 38 and ULOQ = 6960 arbitrary units (AU)/milliliter (mL) for SARS-CoV-2 Omicron XBB.1.5 antibody. 95% CI was calculated based on the t-distribution of the log-transformed values for GM concentration, then back transformed to the original scale for presentation. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 40 | 38 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
AU/mL | 1567.0 [1134.6 to 2164.4] | 1939.7 [1366.0 to 2754.4] | 427.6 [302.9 to 603.7] | 901.0 [655.9 to 1237.6] | 882.0 [630.5 to 1233.9] | 1108.3 [801.9 to 1531.7] | 679.7 [451.4 to 1023.4] | 878.7 [640.1 to 1206.2] | 904.8 [576.5 to 1420.1] | 1083.7 [744.2 to 1578.3]

6. Primary Outcome: Part 2: Geometric Mean Fold-Rise (GMFR) of Antibodies for Influenza at Day 29, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were converted to the ULOQ. LLOQ = 10 and ULOQ = 3620 for Influenza A H1N1 antibody, LLOQ = 10 and ULOQ = 5120 for Influenza A H3N2 antibody, LLOQ = 10 and ULOQ = 1356 for Influenza B/Victoria-lineage antibody, and LLOQ = 10 and ULOQ = 1280 for Influenza B/Yamagata-lineage antibody. 95% CI was calculated based on the t-distribution of the log-transformed values for GMFR values, then back transformed to the original scale for presentation. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 38 | 38 | 37 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
ratio
  Influenza A H1N1 Antibody | 2.6 [1.8 to 3.9] | 3.5 [2.5 to 4.8] | 3.7 [2.6 to 5.2] | 1.8 [1.4 to 2.2] | 2.2 [1.7 to 2.8] | 2.7 [1.9 to 3.9] | 2.0 [1.6 to 2.5] | 1.9 [1.3 to 2.7] | 2.7 [2.0 to 3.7] | 2.3 [1.6 to 3.1] | 2.9 [2.2 to 3.7]
  Influenza A H3N2 Antibody | 2.8 [2.2 to 3.7] | 2.6 [2.1 to 3.3] | 3.4 [2.5 to 4.6] | 1.8 [1.4 to 2.3] | 1.9 [1.6 to 2.4] | 2.3 [1.7 to 3.1] | 2.0 [1.5 to 2.7] | 1.7 [1.4 to 2.1] | 2.3 [1.9 to 2.7] | 1.8 [1.3 to 2.4] | 2.7 [2.2 to 3.3]
  Influenza B/Victoria-lineage Antibody | 1.7 [1.4 to 2.1] | 2.0 [1.5 to 2.6] | 2.4 [1.7 to 3.2] | 1.4 [1.2 to 1.7] | 1.6 [1.3 to 1.9] | 1.7 [1.5 to 2.1] | 2.1 [1.7 to 2.6] | 1.5 [1.2 to 1.8] | 1.5 [1.3 to 1.7] | 1.5 [1.3 to 1.9] | 1.7 [1.4 to 2.1]
  Influenza B/Yamagata-lineage Antibody | 1.7 [1.4 to 2.2] | 2.3 [1.8 to 2.8] | 2.1 [1.7 to 2.7] | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.7] | 1.6 [1.3 to 2.0] | 1.6 [1.4 to 1.9] | 1.3 [1.1 to 1.6] | 1.6 [1.3 to 2.0] | 1.4 [1.2 to 1.8] | 1.6 [1.3 to 1.8]

7. Primary Outcome: Part 2: GMFR of Antibodies for SARS-CoV-2 at Day 29, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Antibody values reported as below the LLOQ are replaced by 0.5 * LLOQ. Values greater than the ULOQ are converted to the ULOQ. LLOQ = 38 and ULOQ = 6960 AU/mL for SARS-CoV-2 Omicron XBB.1.5 antibody. 95% CI was calculated based on the t-distribution of the log-transformed values for GMFR values, then back transformed to the original scale for presentation. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 40 | 38 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
ratio | 5.4 [3.3 to 8.7] | 9.1 [5.4 to 15.2] | 3.3 [2.1 to 5.2] | 5.4 [3.5 to 8.1] | 4.4 [2.9 to 6.9] | 3.6 [2.5 to 5.1] | 4.5 [2.9 to 6.9] | 4.1 [2.9 to 6.0] | 7.1 [4.4 to 11.4] | 8.0 [5.4 to 11.7]

8. Primary Outcome: Part 2: Influenza: Percentage of Participants With Seroconversion, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Seroconversion was defined as a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40 or a pre-vaccination HAI titer ≥1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Baseline to Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 38 | 38 | 37 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
percentage of participants
  Influenza A H1N1 Antibody | 31.6 [17.5 to 48.7] | 50.0 [33.4 to 66.6] | 51.4 [34.4 to 68.1] | 17.9 [7.5 to 33.5] | 31.0 [17.6 to 47.1] | 30.0 [16.6 to 46.5] | 25.6 [13.0 to 42.1] | 17.5 [7.3 to 32.8] | 34.2 [19.6 to 51.4] | 30.3 [15.6 to 48.7] | 35.7 [21.6 to 52.0]
  Influenza A H3N2 Antibody | 42.1 [26.3 to 59.2] | 36.8 [21.8 to 54.0] | 43.2 [27.1 to 60.5] | 12.8 [4.3 to 27.4] | 23.8 [12.1 to 39.5] | 27.5 [14.6 to 43.9] | 23.1 [11.1 to 39.3] | 15.0 [5.7 to 29.8] | 21.1 [9.6 to 37.3] | 21.2 [9.0 to 38.9] | 42.9 [27.7 to 59.0]
  Influenza B/Victoria-lineage Antibody | 15.8 [6.0 to 31.3] | 15.8 [6.0 to 31.3] | 27.0 [13.8 to 44.1] | 7.7 [1.6 to 20.9] | 9.5 [2.7 to 22.6] | 12.5 [4.2 to 26.8] | 23.1 [11.1 to 39.3] | 12.5 [4.2 to 26.8] | 2.6 [0.1 to 13.8] | 9.1 [1.9 to 24.3] | 11.9 [4.0 to 25.6]
  Influenza B/Yamagata-lineage Antibody | 21.1 [9.6 to 37.3] | 26.3 [13.4 to 43.1] | 27.0 [13.8 to 44.1] | 7.7 [1.6 to 20.9] | 9.5 [2.7 to 22.6] | 12.5 [4.2 to 26.8] | 7.7 [1.6 to 20.9] | 17.5 [7.3 to 32.8] | 13.2 [4.4 to 28.1] | 9.1 [1.9 to 24.3] | 4.8 [0.6 to 16.2]

9. Primary Outcome: Part 2: SARS-CoV-2: Percentage of Participants With Seroresponse, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Seroresponse was defined as an increase from below the LLOQ to ≥4 * LLOQ if Baseline neutralizing antibody (nAb) level was < LLOQ, or ≥4-fold rise if Baseline nAb level was ≥ LLOQ. LLOQ = 38 and ULOQ = 6960 AU/mL for SARS-CoV-2 Omicron XBB.1.5 antibody. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Baseline to Day 29
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 40 | 38 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
percentage of participants | 55.0 [38.5 to 70.7] | 57.9 [40.8 to 73.7] | 33.3 [19.1 to 50.2] | 52.4 [36.4 to 68.0] | 47.5 [31.5 to 63.9] | 33.3 [19.1 to 50.2] | 50.0 [33.8 to 66.2] | 44.7 [28.6 to 61.7] | 63.6 [45.1 to 79.6] | 69.0 [52.9 to 82.4]

10. Secondary Outcome: Part 1: GMT of Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below LLOQ were replaced by 0.5 * LLOQ. Values greater than ULOQ were converted to ULOQ. LLOQ = 10 and ULOQ = 640 for Influenza A H1N1 and Influenza A H3N2 antibody, LLOQ = 10 and ULOQ = 320 for Influenza B/ Victoria, and LLOQ = 10 and ULOQ = 640 for Influenza B/Yamagata antibody. 95% CI was calculated based on t-distribution of log-transformed values for GM titer, then back transformed to original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Baseline (Day 1), Day 29, and Day 181
Population: PP Set. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category. Arms based on the applicable vaccine for this Outcome Measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 50 | 50 | 47 | 52 | 51 | 53 | 36 | 50 | 52 | 37 | 51
titer
  Influenza A H1N1 Antibody: Day 1: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 49 | 31 | 50 | 50 | 47 | 52 | 51 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza A H1N1 Antibody: Day 1 | 49.7 [40.4 to 61.1] | 47.5 [36.9 to 61.2] | 55.0 [42.3 to 71.6] | 55.7 [43.3 to 71.6] | 58.2 [46.3 to 73.1] | 41.4 [29.0 to 59.2] | 55.1 [41.1 to 73.9] | 53.1 [39.5 to 71.3] | 39.1 [29.7 to 51.6] | 57.7 [46.1 to 72.4] | 48.3 [38.5 to 60.6] | 61.8 [47.2 to 81.0] | 48.9 [38.8 to 61.7] | 51.4 [38.5 to 68.8] | 57.3 [45.6 to 72.0] | 59.4 [44.2 to 79.7] | 52.7 [40.8 to 68.2] | 58.5 [47.0 to 72.8] | 77.0 [55.9 to 106.1] | 58.5 [44.8 to 76.3]
  Influenza A H1N1 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 48 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza A H1N1 Antibody: Day 29 | 78.4 [60.9 to 100.8] | 85.7 [62.9 to 116.8] | 108.5 [84.0 to 140.1] | 149.3 [107.5 to 207.3] | 95.8 [74.8 to 122.8] | 104.3 [69.4 to 156.8] | 106.0 [81.5 to 137.9] | 139.5 [99.9 to 194.9] | 82.7 [56.3 to 121.3] | 129.1 [99.9 to 166.8] | 114.0 [82.1 to 158.3] | 145.3 [105.1 to 200.9] | 138.2 [101.7 to 187.7] | 126.4 [98.3 to 162.5] | 120.8 [89.7 to 162.6] | 135.9 [101.5 to 181.9] | 177.6 [135.6 to 232.4] | 142.9 [115.1 to 177.3] | 196.7 [138.2 to 280.1] | 150.5 [115.0 to 197.0]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 32 | 36 | 43 | 22 | 44 | 39 | 25 | 42 | 45 | 40 | 44 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  Influenza A H1N1 Antibody: Day 181 | 104.5 [80.1 to 136.3] | 104.7 [74.8 to 146.7] | 99.3 [74.0 to 133.3] | 148.1 [99.2 to 221.1] | 104.3 [77.6 to 140.3] | 145.6 [104.1 to 203.7] | 127.3 [96.2 to 168.5] | 135.3 [102.4 to 178.7] | 104.2 [73.7 to 147.2] | 140.2 [108.9 to 180.5] | 118.4 [88.4 to 158.7] | 140.6 [108.1 to 182.8] | 174.5 [137.5 to 221.5] | 134.5 [104.6 to 173.0] | 147.9 [113.0 to 193.5] | 157.9 [111.4 to 223.8] | 176.3 [134.6 to 230.8] | 132.5 [105.9 to 165.9] | 156.1 [114.5 to 212.9] | 161.2 [121.6 to 213.8]
  Influenza A H3N2 Antibody: Day 1: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 49 | 50 | 47 | 52 | 51 | 53 | 36 | 50 | 52 | 37 | 50
  Influenza A H3N2 Antibody: Day 1 | 34.4 [25.5 to 46.6] | 34.1 [26.5 to 43.9] | 38.9 [29.3 to 51.5] | 30.7 [23.0 to 41.0] | 43.1 [33.9 to 54.9] | 31.7 [22.4 to 44.8] | 29.0 [21.4 to 39.5] | 37.6 [27.4 to 51.5] | 39.6 [28.3 to 55.2] | 32.1 [24.0 to 43.0] | 27.5 [21.3 to 35.5] | 48.3 [34.7 to 67.3] | 43.9 [33.2 to 58.1] | 38.9 [29.9 to 50.6] | 30.0 [23.9 to 37.6] | 36.0 [26.1 to 49.7] | 32.0 [23.4 to 43.9] | 43.0 [31.3 to 59.2] | 34.8 [25.9 to 46.7] | 33.2 [25.3 to 43.4]
  Influenza A H3N2 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza A H3N2 Antibody: Day 29 | 61.8 [45.6 to 83.8] | 67.7 [48.9 to 93.8] | 88.3 [65.7 to 118.6] | 113.2 [77.6 to 165.0] | 90.7 [65.6 to 125.2] | 119.8 [74.9 to 191.7] | 64.8 [47.8 to 87.9] | 103.4 [78.1 to 136.9] | 94.6 [63.8 to 140.2] | 100.6 [75.5 to 134.1] | 64.5 [45.8 to 90.9] | 111.5 [84.8 to 146.7] | 117.8 [83.2 to 166.6] | 105.6 [79.4 to 140.3] | 73.0 [52.9 to 100.8] | 104.8 [70.3 to 156.0] | 116.3 [84.2 to 160.6] | 107.2 [77.7 to 147.8] | 93.8 [66.2 to 132.9] | 110.8 [78.8 to 155.9]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 32 | 36 | 43 | 22 | 44 | 39 | 25 | 42 | 45 | 40 | 44 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  Influenza A H3N2 Antibody: Day 181 | 85.1 [64.2 to 112.9] | 87.2 [63.2 to 120.3] | 116.9 [80.0 to 170.7] | 146.7 [99.3 to 216.9] | 129.8 [96.2 to 175.2] | 196.4 [125.1 to 308.5] | 91.5 [71.5 to 117.0] | 114.2 [81.4 to 160.2] | 107.2 [72.5 to 158.5] | 117.9 [87.1 to 159.6] | 83.2 [64.9 to 106.6] | 111.2 [87.2 to 141.9] | 140.0 [93.9 to 208.6] | 129.4 [99.5 to 168.4] | 102.1 [73.7 to 141.5] | 149.3 [95.1 to 234.2] | 120.8 [87.8 to 166.2] | 145.7 [111.0 to 191.2] | 111.7 [79.7 to 156.7] | 134.1 [98.6 to 182.3]
  Influenza B/Victoria-lineage Antibody: Day 1: number analyzed (Participants) | 51 | 50 | 49 | 44 | 50 | 30 | 53 | 49 | 31 | 50 | 50 | 46 | 52 | 51 | 53 | 36 | 50 | 52 | 36 | 50
  Influenza B/Victoria-lineage Antibody: Day 1 | 55.4 [41.3 to 74.3] | 49.2 [35.8 to 67.8] | 46.7 [34.0 to 64.2] | 46.8 [34.5 to 63.4] | 73.1 [56.4 to 94.7] | 52.2 [36.7 to 74.3] | 72.5 [56.2 to 93.7] | 55.0 [41.3 to 73.0] | 46.8 [32.5 to 67.3] | 69.6 [52.3 to 92.8] | 34.5 [25.7 to 46.4] | 33.1 [23.5 to 46.6] | 31.5 [23.3 to 42.6] | 37.6 [28.5 to 49.6] | 39.0 [29.2 to 52.0] | 34.3 [23.3 to 50.4] | 35.3 [25.1 to 49.5] | 36.9 [28.2 to 48.4] | 33.0 [24.7 to 44.1] | 39.4 [28.6 to 54.4]
  Influenza B/Victoria-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 44 | 50 | 30 | 53 | 48 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza B/Victoria-lineage Antibody: Day 29 | 100.7 [70.1 to 144.8] | 106.3 [72.7 to 155.3] | 88.3 [65.3 to 119.4] | 151.5 [120.5 to 190.5] | 141.2 [107.9 to 184.9] | 128.5 [82.0 to 201.3] | 148.0 [115.3 to 189.9] | 155.5 [121.1 to 199.6] | 152.9 [106.7 to 219.1] | 172.7 [131.9 to 226.0] | 83.4 [58.7 to 118.6] | 59.1 [44.7 to 78.2] | 83.8 [59.7 to 117.6] | 76.8 [59.5 to 99.1] | 96.7 [70.2 to 133.0] | 89.0 [62.1 to 127.7] | 76.1 [55.1 to 105.2] | 113.1 [82.1 to 155.9] | 91.2 [65.2 to 127.7] | 93.5 [67.1 to 130.3]
  Influenza B/Victoria-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 32 | 36 | 43 | 22 | 44 | 39 | 25 | 42 | 45 | 40 | 44 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  Influenza B/Victoria-lineage Antibody: Day 181 | 167.2 [113.6 to 246.2] | 128.2 [86.3 to 190.6] | 95.1 [68.6 to 131.9] | 139.9 [108.0 to 181.1] | 140.6 [106.9 to 184.8] | 178.8 [110.4 to 289.4] | 174.5 [136.2 to 223.6] | 142.5 [101.1 to 200.9] | 183.7 [122.6 to 275.4] | 185.7 [136.2 to 253.1] | 103.2 [77.5 to 137.4] | 81.3 [58.0 to 113.9] | 115.9 [82.1 to 163.6] | 115.9 [86.8 to 154.6] | 126.3 [97.6 to 163.5] | 82.2 [53.0 to 127.5] | 86.0 [64.1 to 115.4] | 93.8 [73.0 to 120.4] | 99.9 [64.2 to 155.6] | 112.3 [81.4 to 155.0]
  Influenza B/Yamagata-lineage Antibody: Day 1: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 50 | 50 | 47 | 52 | 51 | 53 | 36 | 50 | 52 | 37 | 50
  Influenza B/Yamagata-lineage Antibody: Day 1 | 49.0 [36.9 to 65.2] | 56.5 [43.0 to 74.3] | 62.9 [46.5 to 85.0] | 52.7 [39.7 to 70.0] | 80.6 [65.0 to 99.9] | 63.5 [45.3 to 88.9] | 74.5 [57.2 to 96.9] | 56.5 [42.8 to 74.7] | 48.4 [33.1 to 70.7] | 90.6 [68.8 to 119.4] | 78.3 [62.4 to 98.3] | 94.1 [74.0 to 119.6] | 85.5 [66.5 to 110.0] | 100.1 [74.0 to 135.4] | 91.1 [67.9 to 122.2] | 81.6 [60.9 to 109.3] | 74.7 [57.8 to 96.5] | 88.5 [67.6 to 115.8] | 101.1 [71.0 to 143.9] | 84.0 [62.2 to 113.5]
  Influenza B/Yamagata-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 48 | 31 | 50 | 50 | 47 | 52 | 50 | 52 | 36 | 50 | 52 | 37 | 51
  Influenza B/Yamagata-lineage Antibody: Day 29 | 75.2 [56.2 to 100.7] | 110.0 [83.3 to 145.3] | 100.4 [75.9 to 132.8] | 108.1 [82.3 to 141.9] | 110.8 [86.9 to 141.3] | 101.9 [69.0 to 150.4] | 112.3 [83.3 to 151.5] | 98.7 [75.9 to 128.1] | 80.0 [56.5 to 113.3] | 145.2 [109.5 to 192.7] | 151.4 [108.7 to 210.8] | 165.9 [132.4 to 208.0] | 176.7 [129.5 to 241.3] | 185.0 [134.8 to 253.9] | 178.0 [139.7 to 226.7] | 145.3 [100.5 to 210.0] | 154.5 [118.2 to 202.0] | 181.5 [139.6 to 236.1] | 246.1 [175.8 to 344.6] | 154.7 [113.5 to 210.8]
  Influenza B/Yamagata-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 32 | 36 | 43 | 22 | 44 | 39 | 24 | 42 | 45 | 40 | 44 | 43 | 44 | 25 | 43 | 48 | 28 | 45
  Influenza B/Yamagata-lineage Antibody: Day 181 | 94.8 [65.4 to 137.4] | 112.0 [78.2 to 160.5] | 84.5 [56.5 to 126.4] | 98.9 [68.6 to 142.5] | 109.6 [80.9 to 148.4] | 109.6 [71.7 to 167.6] | 98.9 [74.0 to 132.3] | 98.1 [68.4 to 140.9] | 87.3 [53.2 to 143.1] | 121.9 [87.6 to 169.6] | 88.4 [66.6 to 117.3] | 91.8 [69.2 to 121.8] | 121.4 [89.6 to 164.5] | 129.8 [95.6 to 176.1] | 121.4 [91.5 to 161.0] | 75.7 [50.2 to 114.1] | 112.2 [78.5 to 160.4] | 95.2 [72.9 to 124.1] | 111.7 [76.6 to 162.9] | 88.4 [66.6 to 117.5]

11. Secondary Outcome: Part 1: GMT of Antibodies for SARS-CoV-2, as Measured by PsVNA
Description: SARS-CoV-2 strain included BA.4/5 and D614G antibody. Antibody values reported as below LLOQ were replaced by 0.5 * LLOQ. Values greater than ULOQ were converted to ULOQ. LLOQ = 53 and ULOQ = 71376 for SARS-CoV-2 BA.4/5 antibody and LLOQ = 74.1 and ULOQ = 184317 for SARS-CoV-2 D614G antibody. 95% CI was calculated based on t-distribution of log-transformed values for GM titer, then back transformed to original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Baseline (Day 1), Day 29, and Day 181
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 49 | 50 | 30 | 53 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 51
titer
  SARS-CoV-2 BA.4/5 Antibody: Day 1: number analyzed (Participants) | 51 | 49 | 50 | 29 | 52 | 51 | 31 | 50 | 50 | 52 | 51 | 53 | 36 | 50 | 52 | 38 | 51
  SARS-CoV-2 BA.4/5 Antibody: Day 1 | 618.0 [403.0 to 947.9] | 574.1 [352.8 to 848.2] | 616.9 [367.1 to 1036.8] | 585.9 [314.7 to 1090.6] | 646.6 [408.8 to 1022.7] | 536.3 [329.5 to 872.7] | 1008.2 [616.1 to 1649.7] | 883.2 [584.9 to 1333.6] | 384.1 [251.4 to 586.8] | 469.8 [297.5 to 741.8] | 653.7 [442.5 to 965.8] | 440.5 [295.7 to 656.3] | 487.5 [283.4 to 838.4] | 469.1 [292.1 to 753.2] | 524.8 [361.7 to 761.5] | 301.8 [195.0 to 467.1] | 489.8 [320.9 to 747.7]
  SARS-CoV-2 BA.4/5 Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 50 | 30 | 53 | 51 | 31 | 50 | 50 | 52 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 BA.4/5 Antibody: Day 29 | 4536.9 [3147.0 to 6540.8] | 5476.9 [3988.2 to 7521.5] | 4636.7 [3098.6 to 6938.3] | 5387.3 [3207.7 to 9047.8] | 3706.0 [2656.8 to 5169.4] | 3669.6 [2577.8 to 5223.8] | 5647.8 [4227.0 to 7546.2] | 4120.6 [3224.4 to 5265.8] | 2635.8 [1973.8 to 3519.9] | 4743.9 [3529.0 to 6377.1] | 4005.9 [3131.4 to 5124.5] | 3061.1 [2308.3 to 4059.2] | 3599.0 [2577.6 to 5025.1] | 3425.6 [2558.6 to 4586.4] | 4391.3 [3488.0 to 5528.4] | 3119.7 [2360.0 to 4124.0] | 3458.4 [2595.9 to 4607.5]
  SARS-CoV-2 BA.4/5 Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 44 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  SARS-CoV-2 BA.4/5 Antibody: Day 181 | 1500.1 [977.6 to 2301.8] | 2524.4 [1588.3 to 4012.3] | 1793.9 [1145.8 to 2808.5] | 1851.8 [899.5 to 3812.3] | 1461.3 [945.9 to 2257.6] | 1552.5 [935.1 to 2577.6] | 2185.7 [1425.4 to 3351.4] | 1480.3 [980.2 to 2235.6] | 1443.0 [1049.6 to 1983.9] | 1972.1 [1305.9 to 2978.2] | 1595.9 [1167.3 to 2181.8] | 1225.0 [861.6 to 1741.6] | 1657.5 [999.9 to 2747.5] | 1413.4 [936.8 to 2132.5] | 1792.7 [1311.6 to 2450.4] | 1042.8 [620.3 to 1753.1] | 1270.3 [888.8 to 1815.5]
  SARS-CoV-2 D614G Antibody: Day 1: number analyzed (Participants) | 51 | 49 | 50 | 30 | 52 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 D614G Antibody: Day 1 | 2052.1 [1472.4 to 2860.0] | 2176.0 [1546.4 to 3062.0] | 2362.5 [1525.7 to 3658.3] | 2578.4 [1482.4 to 4484.8] | 2992.6 [2118.7 to 4226.9] | 2091.1 [1408.0 to 3105.7] | 3284.9 [2260.6 to 4773.3] | 2909.8 [2255.8 to 3753.4] | 1548.5 [1057.5 to 2267.5] | 1756.8 [1185.2 to 2604.2] | 2328.9 [1776.8 to 3052.6] | 1994.9 [1476.1 to 2696.1] | 1553.2 [1011.9 to 2384.1] | 1575.1 [1051.1 to 2360.4] | 2056.3 [1471.1 to 2874.2] | 1391.3 [986.7 to 1961.7] | 1527.4 [1057.0 to 2207.2]
  SARS-CoV-2 D614G Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 48 | 30 | 53 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 D614G Antibody: Day 29 | 9943.4 [7910.9 to 12498.1] | 12229.6 [9571.1 to 15626.7] | 9275.7 [6926.0 to 12422.7] | 10433.9 [7040.4 to 15463.1] | 7678.3 [6034.4 to 9770.0] | 8513.1 [6542.0 to 11078.0] | 10057.5 [7712.1 to 13116.1] | 8639.7 [7025.9 to 10624.1] | 7038.1 [5592.1 to 8858.0] | 10243.2 [8204.9 to 12787.7] | 7431.1 [6091.6 to 9065.1] | 7127.4 [5855.8 to 8675.1] | 6525.4 [4850.0 to 8779.4] | 6738.9 [5281.8 to 8597.8] | 7844.9 [6467.6 to 9515.4] | 7333.0 [5842.7 to 9203.4] | 6877.4 [5218.1 to 9064.5]
  SARS-CoV-2 D614G Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 44 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  SARS-CoV-2 D614G Antibody: Day 181 | 3583.2 [2756.2 to 4658.4] | 5778.1 [4110.6 to 8121.9] | 4006.2 [2759.3 to 5816.7] | 3927.0 [2086.7 to 7390.1] | 3317.4 [2397.5 to 4590.2] | 3877.3 [2667.2 to 5636.2] | 5622.0 [3718.2 to 8500.5] | 3889.4 [2807.8 to 5387.6] | 3296.0 [2452.4 to 4429.8] | 4324.3 [3256.8 to 5741.6] | 3292.4 [2601.5 to 4166.7] | 3008.6 [2336.9 to 3873.5] | 2633.9 [1532.5 to 4527.0] | 2743.1 [1976.1 to 3807.9] | 2904.4 [2145.9 to 3931.1] | 1908.1 [1316.1 to 2766.3] | 2386.0 [1676.1 to 3396.6]

12. Secondary Outcome: Part 1: GMFR of Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below LLOQ were replaced by 0.5 * LLOQ. Values greater than ULOQ were converted to ULOQ. LLOQ = 10 and ULOQ = 640 for Influenza A H1N1 and Influenza A H3N2 antibody, LLOQ = 10 and ULOQ = 320 for Influenza B/Victoria, and LLOQ = 10 and ULOQ = 640 for Influenza B/Yamagata antibody. 95% CI was calculated based on t-distribution of log-transformed values for GMFR, then back transformed to original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Day 29 and Day 181
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
ratio
  Influenza A H1N1 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 47 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza A H1N1 Antibody: Day 29 | 1.6 [1.2 to 2.0] | 1.8 [1.5 to 2.2] | 2.0 [1.7 to 2.3] | 2.7 [2.0 to 3.6] | 1.6 [1.4 to 2.0] | 2.5 [1.8 to 3.6] | 1.9 [1.5 to 2.4] | 2.6 [2.1 to 3.4] | 2.1 [1.6 to 2.8] | 2.2 [1.7 to 2.9] | 2.4 [1.8 to 3.2] | 2.4 [1.8 to 3.0] | 2.8 [2.1 to 3.9] | 2.4 [1.8 to 3.3] | 2.1 [1.6 to 2.7] | 2.3 [1.8 to 3.0] | 3.4 [2.5 to 4.5] | 2.4 [1.8 to 3.3] | 2.6 [1.7 to 3.8] | 2.6 [2.0 to 3.3]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 37 | 25 | 42 | 45 | 39 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 45
  Influenza A H1N1 Antibody: Day 181 | 2.1 [1.6 to 2.8] | 1.8 [1.3 to 2.4] | 1.8 [1.4 to 2.2] | 2.6 [1.6 to 4.2] | 1.9 [1.5 to 2.3] | 3.6 [2.6 to 5.0] | 2.4 [1.8 to 3.2] | 2.7 [2.0 to 3.7] | 2.6 [1.9 to 3.7] | 2.4 [1.9 to 3.2] | 2.5 [1.8 to 3.4] | 2.4 [1.9 to 3.1] | 3.2 [2.6 to 4.1] | 3.0 [2.2 to 4.1] | 2.3 [1.8 to 3.1] | 3.0 [2.1 to 4.3] | 3.3 [2.5 to 4.3] | 2.3 [1.7 to 3.1] | 2.3 [1.6 to 3.3] | 2.7 [2.0 to 3.6]
  Influenza A H3N2 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 49 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 50
  Influenza A H3N2 Antibody: Day 29 | 1.8 [1.4 to 2.3] | 2.0 [1.6 to 2.5] | 2.3 [1.8 to 2.8] | 3.7 [2.8 to 4.8] | 2.1 [1.7 to 2.6] | 3.8 [2.5 to 5.6] | 2.2 [1.8 to 2.8] | 2.8 [2.1 to 3.6] | 2.4 [1.7 to 3.4] | 3.1 [2.4 to 3.9] | 2.3 [1.8 to 3.0] | 2.3 [1.8 to 2.9] | 2.7 [2.1 to 3.5] | 2.7 [2.0 to 3.7] | 2.4 [1.8 to 3.3] | 2.9 [2.2 to 3.8] | 3.6 [2.6 to 5.0] | 2.5 [1.8 to 3.5] | 2.7 [1.9 to 3.8] | 3.3 [2.6 to 4.2]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 38 | 25 | 41 | 45 | 39 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza A H3N2 Antibody: Day 181 | 2.5 [1.8 to 3.4] | 2.2 [1.6 to 2.9] | 3.2 [2.4 to 4.2] | 4.6 [3.1 to 6.8] | 2.9 [2.3 to 3.5] | 5.7 [3.4 to 9.5] | 3.2 [2.4 to 4.4] | 3.2 [2.3 to 4.3] | 2.7 [1.9 to 3.9] | 3.9 [3.0 to 5.0] | 3.0 [2.3 to 3.9] | 2.6 [1.9 to 3.4] | 3.2 [2.3 to 4.5] | 3.5 [2.5 to 4.8] | 3.5 [2.4 to 5.0] | 4.3 [2.9 to 6.4] | 3.8 [2.6 to 5.8] | 3.2 [2.3 to 4.3] | 3.3 [2.4 to 4.4] | 3.9 [2.8 to 5.5]
  Influenza B/Victoria-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 43 | 50 | 30 | 53 | 47 | 31 | 50 | 50 | 46 | 52 | 50 | 53 | 36 | 50 | 52 | 36 | 50
  Influenza B/Victoria-lineage Antibody: Day 29 | 1.8 [1.3 to 2.5] | 2.2 [1.6 to 2.9] | 1.9 [1.5 to 2.4] | 3.3 [2.4 to 4.6] | 1.9 [1.6 to 2.4] | 2.5 [1.6 to 3.7] | 2.0 [1.7 to 2.4] | 2.9 [2.2 to 3.8] | 3.3 [2.3 to 4.7] | 2.5 [1.9 to 3.3] | 2.4 [1.8 to 3.2] | 1.9 [1.5 to 2.3] | 2.7 [2.1 to 3.4] | 2.1 [1.8 to 2.5] | 2.5 [1.8 to 3.4] | 2.6 [1.9 to 3.6] | 2.2 [1.7 to 2.8] | 3.1 [2.4 to 3.9] | 2.7 [2.0 to 3.8] | 2.4 [1.9 to 3.0]
  Influenza B/Victoria-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 35 | 43 | 22 | 44 | 37 | 25 | 42 | 45 | 38 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza B/Victoria-lineage Antibody: Day 181 | 2.9 [2.1 to 4.0] | 2.4 [1.7 to 3.4] | 2.1 [1.7 to 2.7] | 2.9 [2.0 to 4.3] | 1.9 [1.5 to 2.3] | 3.2 [2.1 to 5.0] | 2.3 [1.8 to 2.8] | 2.4 [1.7 to 3.4] | 4.0 [2.7 to 5.8] | 2.9 [2.2 to 3.9] | 3.1 [2.3 to 4.2] | 2.2 [1.6 to 2.9] | 3.4 [2.6 to 4.6] | 3.1 [2.3 to 4.0] | 3.6 [2.7 to 4.7] | 3.0 [1.8 to 5.0] | 2.5 [1.8 to 3.4] | 2.6 [2.1 to 3.2] | 3.1 [2.0 to 4.6] | 2.9 [2.1 to 4.0]
  Influenza B/Yamagata-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 48 | 31 | 50 | 50 | 47 | 52 | 50 | 52 | 36 | 50 | 52 | 37 | 50
  Influenza B/Yamagata-lineage Antibody: Day 29 | 1.5 [1.2 to 1.9] | 1.9 [1.5 to 2.6] | 1.6 [1.3 to 1.9] | 2.0 [1.6 to 2.6] | 1.4 [1.2 to 1.6] | 1.6 [1.2 to 2.1] | 1.5 [1.2 to 1.8] | 1.8 [1.5 to 2.2] | 1.7 [1.2 to 2.2] | 1.6 [1.3 to 1.9] | 1.9 [1.5 to 2.5] | 1.8 [1.5 to 2.1] | 2.1 [1.6 to 2.7] | 1.9 [1.5 to 2.4] | 2.0 [1.6 to 2.6] | 1.8 [1.4 to 2.2] | 2.1 [1.7 to 2.6] | 2.1 [1.8 to 2.4] | 2.4 [1.8 to 3.3] | 1.9 [1.5 to 2.4]
  Influenza B/Yamagata-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 38 | 24 | 42 | 45 | 39 | 44 | 43 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza B/Yamagata-lineage Antibody: Day 181 | 1.9 [1.3 to 2.7] | 1.8 [1.1 to 3.0] | 1.3 [0.8 to 2.2] | 2.0 [1.3 to 3.0] | 1.3 [1.0 to 1.6] | 1.7 [1.0 to 2.9] | 1.2 [0.9 to 1.7] | 1.6 [1.0 to 2.7] | 2.0 [1.3 to 3.3] | 1.4 [1.0 to 1.9] | 1.1 [0.8 to 1.4] | 0.9 [0.7 to 1.3] | 1.4 [1.0 to 1.9] | 1.3 [0.9 to 1.8] | 1.4 [1.0 to 1.9] | 0.9 [0.7 to 1.3] | 1.5 [1.1 to 2.1] | 1.1 [0.8 to 1.6] | 1.2 [0.9 to 1.8] | 1.1 [0.8 to 1.5]

13. Secondary Outcome: Part 1: GMFR of Antibodies for SARS-CoV-2, as Measured by PsVNA
Description: SARS-CoV-2 strain included BA.4/5 and D614G antibody. Antibody values reported as below LLOQ were replaced by 0.5 * LLOQ. Values greater than ULOQ were converted to ULOQ. LLOQ = 53 and ULOQ = 71376 for SARS-CoV-2 BA.4/5 antibody and LLOQ = 74.1 and ULOQ = 184317 for SARS-CoV-2 D614G antibody. 95% CI was calculated based on t-distribution of log-transformed values for GMFR, then back transformed to original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Day 29 and Day 181
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 49 | 50 | 30 | 52 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
ratio
  SARS-CoV-2 BA.4/5 Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 50 | 29 | 52 | 51 | 31 | 50 | 50 | 51 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 BA.4/5 Antibody: Day 29 | 7.3 [5.0 to 10.9] | 10.0 [7.0 to 14.2] | 7.5 [5.0 to 11.2] | 9.6 [6.5 to 14.4] | 5.7 [4.1 to 7.9] | 6.8 [4.8 to 9.7] | 5.6 [3.7 to 8.5] | 4.7 [3.3 to 6.7] | 6.9 [4.7 to 10.0] | 10.9 [7.5 to 15.9] | 6.1 [4.2 to 9.0] | 6.9 [5.1 to 9.5] | 7.4 [4.9 to 11.1] | 7.3 [5.1 to 10.5] | 8.4 [5.9 to 11.8] | 10.3 [6.7 to 16.0] | 6.9 [4.6 to 10.4]
  SARS-CoV-2 BA.4/5 Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 43 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  SARS-CoV-2 BA.4/5 Antibody: Day 181 | 2.5 [1.7 to 3.6] | 4.1 [2.7 to 6.3] | 3.2 [2.1 to 5.0] | 4.4 [2.3 to 8.4] | 2.6 [1.8 to 3.8] | 2.4 [1.6 to 3.8] | 1.9 [1.1 to 3.2] | 1.7 [1.1 to 2.5] | 3.5 [2.2 to 5.5] | 4.4 [3.1 to 6.4] | 2.8 [1.9 to 4.1] | 2.7 [1.9 to 3.9] | 2.7 [1.5 to 4.6] | 3.1 [2.1 to 4.6] | 3.5 [2.4 to 5.0] | 3.6 [2.4 to 5.3] | 2.9 [2.0 to 4.3]
  SARS-CoV-2 D614G Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 48 | 30 | 52 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 D614G Antibody: Day 29 | 4.8 [3.6 to 6.5] | 5.6 [4.1 to 7.7] | 4.2 [2.9 to 6.0] | 4.0 [2.9 to 5.6] | 2.5 [1.9 to 3.4] | 4.1 [2.9 to 5.7] | 3.1 [2.2 to 4.2] | 3.0 [2.4 to 3.7] | 4.5 [3.4 to 6.2] | 5.8 [4.0 to 8.5] | 3.2 [2.4 to 4.2] | 3.6 [2.7 to 4.7] | 4.2 [3.1 to 5.7] | 4.3 [3.1 to 5.9] | 3.8 [2.9 to 5.1] | 5.3 [3.8 to 7.3] | 4.5 [3.2 to 6.3]
  SARS-CoV-2 D614G Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 43 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 44
  SARS-CoV-2 D614G Antibody: Day 181 | 1.7 [1.3 to 2.3] | 2.5 [1.7 to 3.8] | 1.7 [1.1 to 2.4] | 1.6 [1.0 to 2.8] | 1.2 [0.9 to 1.6] | 1.7 [1.2 to 2.4] | 1.6 [1.1 to 2.4] | 1.4 [1.1 to 1.7] | 2.0 [1.3 to 2.9] | 2.5 [1.8 to 3.5] | 1.5 [1.2 to 1.8] | 1.5 [1.1 to 2.1] | 1.4 [1.1 to 1.9] | 1.7 [1.3 to 2.3] | 1.4 [1.0 to 1.9] | 1.5 [1.2 to 2.0] | 1.7 [1.2 to 2.4]

14. Secondary Outcome: Part 1: Influenza: Percentage of Participants With Seroconversion, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Seroconversion was defined as a pre-vaccination HAI titer < 1:10 and a post-vaccination HAI titer ≥1:40 or a pre-vaccination HAI titer ≥1:10 and a minimum 4-fold rise in post vaccination HAI antibody titer. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Baseline (Day 1) to Day 29, and Day 181
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
percentage of participants
  Influenza A H1N1 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 47 | 31 | 50 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 51
  Influenza A H1N1 Antibody: Day 29 | 11.8 [4.4 to 23.9] | 14.0 [5.8 to 26.7] | 18.4 [8.8 to 32.0] | 28.9 [16.4 to 44.3] | 12.0 [4.5 to 24.3] | 33.3 [17.3 to 52.8] | 20.8 [10.8 to 34.1] | 34.0 [20.9 to 49.3] | 19.4 [7.5 to 37.5] | 18.0 [8.6 to 31.4] | 30.0 [17.9 to 44.6] | 27.7 [15.6 to 42.6] | 36.5 [23.6 to 51.0] | 30.0 [17.9 to 44.6] | 20.8 [10.8 to 34.1] | 19.4 [8.2 to 36.0] | 48.0 [33.7 to 62.6] | 30.8 [18.7 to 45.1] | 29.7 [15.9 to 47.0] | 37.3 [24.1 to 51.9]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 37 | 25 | 42 | 45 | 39 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 45
  Influenza A H1N1 Antibody: Day 181 | 28.2 [15.0 to 44.9] | 16.7 [6.4 to 32.8] | 16.1 [5.5 to 33.7] | 30.6 [16.3 to 48.1] | 23.3 [11.8 to 38.6] | 50.0 [28.2 to 71.8] | 27.3 [15.0 to 42.8] | 32.4 [18.0 to 49.8] | 36.0 [18.0 to 57.5] | 21.4 [10.3 to 36.8] | 31.1 [18.2 to 46.6] | 33.3 [19.1 to 50.2] | 40.9 [26.3 to 56.8] | 40.9 [26.3 to 56.8] | 38.6 [24.4 to 54.5] | 36.0 [18.0 to 57.5] | 44.2 [29.1 to 60.1] | 29.2 [17.0 to 44.1] | 29.6 [13.8 to 50.2] | 37.8 [23.8 to 53.5]
  Influenza A H3N2 Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 50 | 31 | 49 | 50 | 47 | 52 | 50 | 53 | 36 | 50 | 52 | 37 | 50
  Influenza A H3N2 Antibody: Day 29 | 15.7 [7.0 to 28.6] | 22.0 [11.5 to 36.0] | 22.4 [11.8 to 36.6] | 55.6 [40.0 to 70.4] | 26.0 [14.6 to 40.3] | 43.3 [25.5 to 62.6] | 22.6 [12.3 to 36.2] | 38.0 [24.7 to 52.8] | 25.8 [11.9 to 44.6] | 44.9 [30.7 to 59.8] | 32.0 [19.5 to 46.7] | 31.9 [19.1 to 47.1] | 40.4 [27.0 to 54.9] | 34.0 [21.2 to 48.8] | 24.5 [13.8 to 38.3] | 44.4 [27.9 to 61.9] | 44.0 [30.0 to 58.7] | 38.5 [25.3 to 53.0] | 35.1 [20.2 to 52.5] | 34.0 [21.2 to 48.8]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 38 | 25 | 41 | 45 | 39 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza A H3N2 Antibody: Day 181 | 33.3 [19.1 to 50.2] | 25.0 [12.1 to 42.2] | 45.2 [27.3 to 64.0] | 61.1 [43.5 to 76.9] | 39.5 [25.0 to 55.6] | 63.6 [40.7 to 82.8] | 43.2 [28.3 to 59.0] | 50.0 [33.4 to 66.6] | 32.0 [14.9 to 53.5] | 51.2 [35.1 to 67.1] | 44.4 [29.6 to 60.0] | 30.8 [17.0 to 47.6] | 47.7 [32.5 to 63.3] | 38.6 [24.4 to 54.5] | 38.6 [24.4 to 54.5] | 44.0 [24.4 to 65.1] | 46.5 [31.2 to 62.3] | 52.1 [37.2 to 66.7] | 40.7 [22.4 to 61.2] | 52.3 [36.7 to 67.5]
  Influenza B/Victoria-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 43 | 50 | 30 | 53 | 47 | 31 | 50 | 50 | 46 | 52 | 50 | 53 | 36 | 50 | 52 | 36 | 50
  Influenza B/Victoria-lineage Antibody: Day 29 | 21.6 [11.3 to 35.3] | 18.0 [8.6 to 31.4] | 22.4 [11.8 to 36.6] | 48.8 [33.3 to 64.5] | 16.0 [7.2 to 29.1] | 23.3 [9.9 to 42.3] | 24.5 [13.8 to 38.3] | 36.2 [22.7 to 51.5] | 41.9 [24.5 to 60.9] | 28.0 [16.2 to 42.5] | 34.0 [21.2 to 48.8] | 13.0 [4.9 to 26.3] | 38.5 [25.3 to 53.0] | 16.0 [7.2 to 29.1] | 34.0 [21.5 to 48.3] | 38.9 [23.1 to 56.5] | 28.0 [16.2 to 42.5] | 38.5 [25.3 to 53.0] | 38.9 [23.1 to 56.5] | 28.0 [16.2 to 42.5]
  Influenza B/Victoria-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 35 | 43 | 22 | 44 | 37 | 25 | 42 | 45 | 38 | 44 | 44 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza B/Victoria-lineage Antibody: Day 181 | 35.9 [21.2 to 52.8] | 27.8 [14.2 to 45.2] | 25.8 [11.9 to 44.6] | 37.1 [21.5 to 55.1] | 18.6 [8.4 to 33.4] | 50.0 [28.2 to 71.8] | 20.5 [9.8 to 35.3] | 32.4 [18.0 to 49.8] | 60.0 [38.7 to 78.9] | 33.3 [19.6 to 49.5] | 48.9 [33.7 to 64.2] | 31.6 [17.5 to 48.7] | 43.2 [28.3 to 59.0] | 47.7 [32.5 to 63.3] | 45.5 [30.4 to 61.2] | 32.0 [14.9 to 53.5] | 32.6 [19.1 to 48.5] | 35.4 [22.2 to 50.5] | 48.1 [28.7 to 68.1] | 45.5 [30.4 to 61.2]
  Influenza B/Yamagata-lineage Antibody: Day 29: number analyzed (Participants) | 51 | 50 | 49 | 45 | 50 | 30 | 53 | 48 | 31 | 50 | 50 | 47 | 52 | 50 | 52 | 36 | 50 | 52 | 37 | 50
  Influenza B/Yamagata-lineage Antibody: Day 29 | 9.8 [3.3 to 21.4] | 18.0 [8.6 to 31.4] | 12.2 [4.6 to 24.8] | 28.9 [16.4 to 44.3] | 2.0 [0.1 to 10.6] | 13.3 [3.8 to 30.7] | 7.5 [2.1 to 18.2] | 16.7 [7.5 to 30.2] | 16.1 [5.5 to 33.7] | 6.0 [1.3 to 16.5] | 24.0 [13.1 to 38.2] | 12.8 [4.8 to 25.7] | 23.1 [12.5 to 36.8] | 20.0 [10.0 to 33.7] | 21.2 [11.1 to 34.7] | 19.4 [8.2 to 36.0] | 20.0 [10.0 to 33.7] | 17.3 [8.2 to 30.3] | 32.4 [18.0 to 49.8] | 16.0 [7.2 to 29.1]
  Influenza B/Yamagata-lineage Antibody: Day 181: number analyzed (Participants) | 39 | 36 | 31 | 36 | 43 | 22 | 44 | 38 | 24 | 42 | 45 | 39 | 44 | 43 | 44 | 25 | 43 | 48 | 27 | 44
  Influenza B/Yamagata-lineage Antibody: Day 181 | 28.2 [15.0 to 44.9] | 33.3 [18.6 to 51.0] | 19.4 [7.5 to 37.5] | 36.1 [20.8 to 53.8] | 9.3 [2.6 to 22.1] | 27.3 [10.7 to 50.2] | 15.9 [6.6 to 30.1] | 23.7 [11.4 to 40.2] | 29.2 [12.6 to 51.1] | 19.0 [8.6 to 34.1] | 8.9 [2.5 to 21.2] | 12.8 [4.3 to 27.4] | 18.2 [8.2 to 32.7] | 20.9 [10.0 to 36.0] | 15.9 [6.6 to 30.1] | 0 [0.0 to 13.7] | 16.3 [6.8 to 30.7] | 14.6 [6.1 to 27.8] | 14.8 [4.2 to 33.7] | 11.4 [3.8 to 24.6]

15. Secondary Outcome: Part 1: SARS-CoV-2: Percentage of Participants With Seroresponse, as Measured by PsVNA
Description: SARS-CoV-2 strain included BA.4/5 and D614G antibody. Seroresponse was defined as an increase from below the LLOQ to ≥4 x LLOQ if baseline nAb level was <LLOQ, or ≥4 fold rise if baseline nAb level was ≥LLOQ. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Baseline (Day 1) to Day 29, and Day 181
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3
Number analyzed (Participants) | 51 | 49 | 50 | 30 | 52 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
percentage of participants
  SARS-CoV-2 BA.4/5 Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 50 | 29 | 52 | 51 | 31 | 50 | 50 | 51 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 BA.4/5 Antibody: Day 29 | 62.7 [48.1 to 75.9] | 69.4 [54.6 to 81.7] | 68.0 [53.3 to 80.5] | 75.9 [56.5 to 89.7] | 56.9 [45.1 to 73.0] | 62.7 [48.1 to 75.9] | 58.1 [39.1 to 75.5] | 44.0 [30.0 to 58.7] | 60.0 [45.2 to 73.6] | 76.5 [62.5 to 87.2] | 51.0 [36.6 to 65.2] | 62.3 [47.9 to 75.5] | 58.3 [40.8 to 74.5] | 60.0 [45.2 to 73.6] | 65.4 [50.9 to 78.0] | 68.4 [51.3 to 82.5] | 68.0 [53.3 to 80.5]
  SARS-CoV-2 BA.4/5 Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 43 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 45
  SARS-CoV-2 BA.4/5 Antibody: Day 181 | 37.8 [23.8 to 53.5] | 44.7 [28.6 to 61.7] | 41.9 [27.0 to 57.9] | 50.0 [28.2 to 71.8] | 41.9 [27.0 to 57.9] | 28.2 [15.0 to 44.9] | 20.0 [6.8 to 40.7] | 16.7 [7.0 to 31.4] | 40.9 [26.3 to 56.8] | 53.2 [38.1 to 67.9] | 29.5 [16.8 to 45.2] | 31.8 [18.6 to 47.6] | 32.0 [14.9 to 53.5] | 34.9 [21.0 to 50.9] | 39.6 [25.8 to 54.7] | 42.9 [24.5 to 62.8] | 35.6 [21.9 to 51.2]
  SARS-CoV-2 D614G Antibody: Day 29: number analyzed (Participants) | 51 | 49 | 48 | 30 | 52 | 51 | 31 | 50 | 50 | 53 | 51 | 53 | 36 | 50 | 52 | 38 | 50
  SARS-CoV-2 D614G Antibody: Day 29 | 43.1 [29.3 to 57.8] | 57.1 [42.2 to 71.2] | 37.5 [24.0 to 52.6] | 56.7 [37.4 to 74.5] | 21.2 [11.1 to 34.7] | 43.1 [29.3 to 57.8] | 25.8 [11.9 to 44.6] | 32.0 [19.5 to 46.7] | 42.0 [28.2 to 56.8] | 50.9 [36.8 to 64.9] | 33.3 [20.8 to 47.9] | 39.6 [26.5 to 54.0] | 41.7 [25.5 to 59.2] | 42.0 [28.2 to 56.8] | 48.1 [34.0 to 62.4] | 57.9 [40.8 to 73.7] | 42.0 [28.2 to 56.8]
  SARS-CoV-2 D614G Antibody: Day 181: number analyzed (Participants) | 45 | 38 | 43 | 22 | 43 | 39 | 25 | 42 | 44 | 47 | 44 | 44 | 25 | 43 | 48 | 28 | 44
  SARS-CoV-2 D614G Antibody: Day 181 | 17.8 [8.0 to 32.1] | 31.6 [17.5 to 48.7] | 18.6 [8.4 to 33.4] | 18.2 [5.2 to 40.3] | 7.0 [1.5 to 19.1] | 17.9 [7.5 to 33.5] | 12.0 [2.5 to 31.2] | 7.1 [1.5 to 19.5] | 22.7 [11.5 to 37.8] | 34.0 [20.9 to 49.3] | 9.1 [2.5 to 21.7] | 11.4 [3.8 to 24.6] | 8.0 [1.0 to 26.0] | 23.3 [11.8 to 38.6] | 12.5 [4.7 to 25.2] | 3.6 [0.1 to 18.3] | 15.9 [6.6 to 30.1]

16. Secondary Outcome: Part 2: GMT of Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were converted to the ULOQ. LLOQ = 10 and ULOQ = 3620 for Influenza A H1N1 antibody, LLOQ = 10 and ULOQ = 5120 for Influenza A H3N2 antibody, LLOQ = 10 and ULOQ = 1356 for Influenza B/Victoria-lineage antibody, and LLOQ = 10 and ULOQ = 1280 for Influenza B/Yamagata-lineage antibody. 95% CI was calculated based on the t-distribution of the log-transformed values for GM titer, then back transformed to the original scale for presentation. Arms based on the applicable vaccine for this Outcome Measure.
Time Frame: Baseline (Day 1), Day 181
Population: PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 38 | 38 | 37 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
titer
  Influenza A H1N1 Antibody: Day 1 | 30.4 [20.3 to 45.4] | 30.1 [20.7 to 43.9] | 35.1 [24.0 to 51.3] | 41.8 [31.5 to 64.1] | 44.9 [31.5 to 64.1] | 40.6 [29.6 to 55.7] | 49.9 [33.3 to 74.8] | 45.5 [32.6 to 63.5] | 32.7 [22.9 to 46.8] | 31.4 [21.0 to 46.9] | 37.1 [26.7 to 51.6]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
  Influenza A H1N1 Antibody: Day 181 | 81.6 [57.6 to 115.8] | 91.3 [65.4 to 127.6] | 108.4 [74.6 to 157.5] | 95.1 [65.9 to 137.1] | 93.1 [63.1 to 137.4] | 119.9 [87.7 to 163.9] | 111.9 [72.1 to 173.6] | 76.4 [52.4 to 111.4] | 108.4 [78.2 to 150.2] | 82.8 [60.6 to 113.2] | 101.5 [73.1 to 141.1]
  Influenza A H3N2 Antibody: Day 1 | 28.8 [21.3 to 38.8] | 36.5 [24.3 to 54.7] | 46.0 [31.9 to 66.3] | 37.2 [27.8 to 49.8] | 36.8 [28.1 to 48.3] | 46.4 [33.2 to 64.8] | 39.6 [28.9 to 54.4] | 36.6 [26.8 to 50.0] | 35.2 [25.7 to 48.3] | 42.1 [30.5 to 58.3] | 30.2 [22.9 to 39.7]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
  Influenza A H3N2 Antibody: Day 181 | 50.9 [37.1 to 69.8] | 65.2 [45.5 to 93.5] | 100.7 [72.9 to 139.2] | 64.1 [46.3 to 88.8] | 52.6 [38.2 to 72.5] | 89.8 [62.2 to 129.6] | 61.7 [43.7 to 87.0] | 49.3 [35.6 to 68.3] | 63.0 [45.5 to 87.3] | 82.9 [57.6 to 119.2] | 52.4 [37.7 to 72.9]
  Influenza B/Victoria-lineage Antibody: Day 1 | 49.8 [38.6 to 64.2] | 41.0 [31.7 to 53.0] | 60.4 [49.9 to 73.1] | 52.6 [40.7 to 68.0] | 64.6 [49.0 to 85.0] | 62.3 [49.1 to 79.0] | 50.8 [39.0 to 66.2] | 66.1 [49.1 to 89.0] | 53.6 [41.1 to 69.8] | 49.3 [38.3 to 63.5] | 48.7 [37.4 to 63.5]
  Influenza B/Victoria-lineage Antibody: Day 181: number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
  Influenza B/Victoria-lineage Antibody: Day 181 | 54.2 [39.7 to 74.1] | 55.4 [42.4 to 72.5] | 64.9 [47.9 to 87.9] | 56.5 [43.0 to 74.3] | 73.0 [54.6 to 97.4] | 69.9 [51.9 to 94.0] | 71.0 [53.2 to 94.8] | 62.5 [46.7 to 83.7] | 56.0 [44.5 to 70.4] | 62.0 [48.4 to 79.4] | 56.6 [44.8 to 71.4]
  Influenza B/Yamagata-lineage Antibody: Day 1 | 80.8 [60.1 to 108.5] | 54.5 [40.8 to 72.9] | 84.7 [63.7 to 112.6] | 63.0 [47.2 to 83.9] | 70.1 [54.7 to 89.8] | 69.7 [53.6 to 90.5] | 69.4 [52.1 to 92.3] | 72.1 [53.8 to 96.6] | 73.6 [52.3 to 103.6] | 67.6 [49.9 to 91.5] | 63.0 [49.6 to 80.0]
  Influenza B/Yamagata-lineage Antibody: Day 181: number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
  Influenza B/Yamagata-lineage Antibody: Day 181 | 110.8 [82.9 to 148.0] | 92.3 [71.4 to 119.2] | 108.5 [78.7 to 149.4] | 68.5 [50.7 to 92.7] | 70.8 [54.7 to 91.6] | 80.7 [60.9 to 107.0] | 82.6 [59.1 to 115.5] | 60.8 [45.1 to 82.1] | 73.3 [54.0 to 99.6] | 84.7 [63.4 to 113.3] | 63.0 [46.1 to 86.1]

17. Secondary Outcome: Part 2: GM Concentration of Antibodies for SARS-CoV-2, as Measured by PsVNA
Description: as for outcome 5
Time Frame: Baseline (Day 1), Day 181
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 40 | 38 | 39 | 42 | 40 | 39 | 40 | 38 | 33 | 42
AU/mL
  SARS-CoV-2 Omicron XBB.1.5 Antibody: Day 1 | 292.2 [197.1 to 433.1] | 214.1 [145.3 to 315.4] | 128.8 [82.4 to 201.3] | 168.1 [110.3 to 256.1] | 198.5 [121.2 to 325.1] | 307.8 [194.8 to 486.4] | 151.5 [96.2 to 238.6] | 212.0 [140.8 to 319.2] | 127.6 [81.4 to 200.1] | 136.2 [92.0 to 201.7]
  SARS-CoV-2 Omicron XBB.1.5 Antibody: Day 181: number analyzed (Participants) | 37 | 30 | 36 | 34 | 35 | 32 | 38 | 32 | 30 | 32
  SARS-CoV-2 Omicron XBB.1.5 Antibody: Day 181 | 906.7 [678.5 to 1211.6] | 998.7 [640.6 to 1557.2] | 377.8 [258.0 to 553.4] | 562.2 [364.2 to 867.8] | 629.8 [419.3 to 946.0] | 809.5 [555.1 to 1180.3] | 349.0 [225.7 to 539.8] | 642.9 [445.3 to 928.2] | 682.7 [429.1 to 1086.2] | 472 [307.2 to 725.3]

18. Secondary Outcome: Part 2: GMFR of Antibodies for Influenza, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Antibody values reported as below LLOQ replaced by 0.5 * LLOQ. Values greater than ULOQ converted to ULOQ. LLOQ= 10, ULOQ= 3620 for Influenza A H1N1, LLOQ= 10, ULOQ= 5120 for Influenza A H3N2, LLOQ= 10, ULOQ= 1356 for Influenza B/Victoria-lineage, and LLOQ= 10, ULOQ= 1280 for Influenza B/Yamagata-lineage. 95% CI was calculated based on t-distribution of log-transformed values for GMFR, then back transformed to original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Day 181
Population: PP Set. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Arms based on the applicable vaccine for this Outcome Measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
ratio
  Influenza A H1N1 Antibody | 2.9 [2.0 to 4.2] | 3.2 [2.3 to 4.4] | 3.1 [2.2 to 4.3] | 2.3 [1.8 to 2.8] | 2.1 [1.5 to 2.9] | 2.9 [2.2 to 3.9] | 2.3 [1.7 to 3.2] | 1.7 [1.2 to 2.4] | 3.7 [2.4 to 5.6] | 2.8 [2.0 to 4.1] | 3.0 [2.2 to 4.1]
  Influenza A H3N2 Antibody | 2.0 [1.5 to 2.6] | 1.9 [1.5 to 2.6] | 2.1 [1.5 to 2.8] | 1.7 [1.3 to 2.2] | 1.4 [1.0 to 1.8] | 2.0 [1.6 to 2.6] | 1.4 [1.0 to 2.0] | 1.4 [1.1 to 1.7] | 2.0 [1.6 to 2.6] | 1.8 [1.4 to 2.5] | 1.8 [1.4 to 2.5]
  Influenza B/Victoria-lineage Antibody | 1.2 [0.9 to 1.6] | 1.4 [1.1 to 1.9] | 1.1 [0.9 to 1.5] | 1.1 [0.8 to 1.4] | 1.1 [0.8 to 1.5] | 1.2 [0.9 to 1.5] | 1.4 [1.1 to 1.8] | 1.0 [0.7 to 1.3] | 1.2 [0.9 to 1.5] | 1.3 [1.0 to 1.7] | 1.2 [0.9 to 1.5]
  Influenza B/Yamagata-lineage Antibody | 1.3 [1.1 to 1.6] | 1.6 [1.3 to 1.9] | 1.3 [1.0 to 1.6] | 1.1 [0.9 to 1.4] | 1.0 [0.8 to 1.3] | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.6] | 0.9 [0.7 to 1.0] | 1.2 [0.9 to 1.6] | 1.2 [1.0 to 1.6] | 1.1 [0.8 to 1.3]

19. Secondary Outcome: Part 2: GMFR of Antibodies for SARS-CoV-2, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Antibody values reported as below the LLOQ are replaced by 0.5 * LLOQ. Values greater than the ULOQ are converted to the ULOQ. LLOQ = 38 and ULOQ = 6960 AU/mL for SARS-CoV-2 Omicron XBB.1.5 antibody. 95% CI was calculated based on the t-distribution of the log-transformed values for GMFR values, then back transformed to the original scale for presentation. PP Set: all randomized participants who received study drug, complied with injection schedule, complied with timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected immune response.
Time Frame: Day 181
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 37 | 30 | 36 | 34 | 35 | 32 | 38 | 32 | 30 | 32
ratio | 3.3 [2.2 to 4.8] | 4.5 [2.7 to 7.7] | 2.8 [1.8 to 4.5] | 3.7 [2.2 to 6.2] | 3.4 [2.3 to 5.1] | 2.3 [1.5 to 3.5] | 2.5 [1.6 to 4.0] | 2.9 [1.9 to 4.5] | 4.7 [2.7 to 8.1] | 3.9 [2.8 to 5.5]

20. Secondary Outcome: Part 2: Influenza: Percentage of Participants With Seroconversion, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Victoria-lineage and Yamagata-lineage. Seroconversion was defined as a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40 or a pre-vaccination HAI titer ≥1:10 and a minimum 4-fold rise in post-vaccination HAI antibody titer. PP Set included all randomized participants who received the study intervention, complied with the injection schedule, complied with the timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Baseline (Day 1) to Day 181
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 33 | 34 | 33 | 36 | 34 | 36 | 32 | 38 | 32 | 30 | 32
percentage of participants
  Influenza A H1N1 Antibody | 45.5 [28.1 to 63.6] | 50.0 [32.4 to 67.6] | 36.4 [20.4 to 54.9] | 22.2 [10.1 to 39.2] | 23.5 [10.7 to 41.2] | 36.1 [20.8 to 53.8] | 25.0 [11.5 to 43.4] | 26.3 [13.4 to 43.1] | 40.6 [23.7 to 59.4] | 40.0 [22.7 to 59.4] | 43.8 [26.4 to 62.3]
  Influenza A H3N2 Antibody | 30.3 [15.6 to 48.7] | 29.4 [15.1 to 47.5] | 24.2 [11.1 to 42.3] | 19.4 [8.2 to 36.0] | 11.8 [3.3 to 27.5] | 25.0 [12.1 to 42.2] | 15.6 [5.3 to 32.8] | 10.5 [2.9 to 24.8] | 34.4 [18.6 to 53.2] | 26.7 [12.3 to 45.9] | 28.1 [13.7 to 46.7]
  Influenza B/Victoria-lineage Antibody | 12.1 [3.4 to 28.2] | 8.8 [1.9 to 23.7] | 9.1 [1.9 to 24.3] | 5.6 [0.7 to 18.7] | 8.8 [1.9 to 23.7] | 5.6 [0.7 to 18.7] | 9.4 [2.0 to 25.0] | 10.5 [2.9 to 24.8] | 12.5 [3.5 to 29.0] | 10.0 [2.1 to 26.5] | 6.3 [0.8 to 20.8]
  Influenza B/Yamagata-lineage Antibody | 9.1 [1.9 to 24.3] | 8.8 [1.9 to 23.7] | 6.1 [0.7 to 20.2] | 5.6 [0.7 to 18.7] | 2.9 [0.1 to 15.3] | 2.8 [0.1 to 14.5] | 9.4 [2.0 to 25.0] | 2.6 [0.1 to 13.8] | 6.3 [0.8 to 20.8] | 6.7 [0.8 to 20.8] | 0 [0.0 to 10.9]

21. Secondary Outcome: Part 2: SARS-CoV-2: Percentage of Participants With Seroresponse, as Measured by PsVNA
Description: SARS-CoV-2 strain included Omicron XBB.1.5 antibody. Seroresponse was defined as an increase from below the LLOQ to ≥4 * LLOQ if Baseline nAb level was < LLOQ, or ≥4-fold rise if Baseline nAb level was ≥ LLOQ. PP Set included all randomized participants who received the study intervention, complied with the injection schedule, complied with the timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29, had no documented infection of either influenza or SARS-CoV-2 on Day 1 and up to Day 29, had no major dosing error, and had no major protocol deviations or conditions/medications that affected the immune response.
Time Frame: Baseline (Day 1) to Day 181
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
Number analyzed (Participants) | 37 | 30 | 36 | 34 | 35 | 32 | 38 | 32 | 30 | 32
percentage of participants | 40.5 [24.8 to 57.9] | 43.3 [25.5 to 62.6] | 36.1 [20.8 to 53.8] | 32.4 [17.4 to 50.5] | 37.1 [21.5 to 55.1] | 25.0 [11.5 to 43.4] | 31.6 [17.5 to 48.7] | 28.1 [13.7 to 46.7] | 50.0 [31.3 to 68.7] | 50.0 [31.9 to 68.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs, AESIs, MAAEs, and AEs leading to study discontinuation were collected up to Day 181. Other (non-serious) adverse events were collected from the time of injection through 28 days after the injection, unless they met the criteria for AESIs, MAAEs, or AEs led to study discontinuation.
Description: The Safety Set included all randomized participants who received the study intervention. Participants were included in the vaccination group corresponding to what they actually received (as treated).
Arm/Group | Part 1 Cohort A12: Influenza Vaccine 1 | Part 1 Cohort A13: Influenza Vaccine 2 | Part 1 Cohort A11: Investigational Influenza Vaccine 2 | Part 1 Cohort A8: Investigational Influenza Vaccine 1 | Part 1 Cohort A10: COVID-19 Vaccine 1 | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort A7: mRNA-1083.3 | Part 1 Cohort B12: Influenza Vaccine 1 | Part 1 Cohort B11: Investigational Influenza Vaccine 2 | Part 1 Cohort B8: Investigational Influenza Vaccine 1 | Part 1 Cohort B10: COVID-19 Vaccine 1 | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 | Part 1 Cohort B7: mRNA-1083.3 | Part 2: Influenza Vaccine 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 | Part 2: COVID-19 Vaccine 2 | Part 2: Investigational COVID-19 Vaccine 2 | Part 2: mRNA-1083 Composition 1 Dose Level 1 | Part 2: mRNA-1083 Composition 1 Dose Level 2 | Part 2: mRNA-1083 Composition 1 Dose Level 3 | Part 2: mRNA-1083 Composition 1 Dose Level 4 | Part 2: mRNA-1083 Composition 2 Dose Level 1 | Part 2: mRNA-1083 Composition 2 Dose Level 2 | Part 2: mRNA-1083 Composition 2 Dose Level 3 | Part 2: mRNA-1083 Composition 2 Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53 | 0/54 | 0/53 | 0/54 | 0/52 | 0/52 | 0/33 | 0/54 | 0/54 | 0/33 | 0/53 | 0/52 | 0/56 | 0/56 | 0/56 | 0/55 | 0/56 | 0/56 | 0/37 | 0/55 | 0/56 | 0/38 | 0/56 | 0/41 | 0/40 | 0/40 | 0/42 | 0/40 | 0/40 | 0/42 | 0/42 | 0/41 | 0/40 | 0/40 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/54 | 2/53 | 1/54 | 1/51 | 2/54 | 1/52 | 2/51 | 0/33 | 1/55 | 1/53 | 1/33 | 1/53 | 1/52 | 2/55 | 1/55 | 0/53 | 0/55 | 1/56 | 0/55 | 1/37 | 1/56 | 0/54 | 1/38 | 2/54 | 1/40 | 1/39 | 1/40 | 0/42 | 0/40 | 1/40 | 0/42 | 1/41 | 0/41 | 0/40 | 0/40 | 1/40 | 0/42
Other Adverse Events (participants affected / at risk) | 1/54 | 3/53 | 4/54 | 3/51 | 1/54 | 6/52 | 3/51 | 2/33 | 0/55 | 6/53 | 0/33 | 0/53 | 1/52 | 3/55 | 2/55 | 2/53 | 2/55 | 7/56 | 1/55 | 2/37 | 4/56 | 8/54 | 5/38 | 2/54 | 2/40 | 0/39 | 2/40 | 0/42 | 3/40 | 3/40 | 1/42 | 5/41 | 1/41 | 5/40 | 2/40 | 4/40 | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort A12: Influenza Vaccine 1 (N=54) | Part 1 Cohort A13: Influenza Vaccine 2 (N=53) | Part 1 Cohort A11: Investigational Influenza Vaccine 2 (N=54) | Part 1 Cohort A8: Investigational Influenza Vaccine 1 (N=51) | Part 1 Cohort A10: COVID-19 Vaccine 1 (N=54) | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 (N=52) | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 (N=51) | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 (N=33) | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 (N=55) | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 (N=53) | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 (N=33) | Part 1 Cohort A7: mRNA-1083.3 (N=53) | Part 1 Cohort B12: Influenza Vaccine 1 (N=52) | Part 1 Cohort B11: Investigational Influenza Vaccine 2 (N=55) | Part 1 Cohort B8: Investigational Influenza Vaccine 1 (N=55) | Part 1 Cohort B10: COVID-19 Vaccine 1 (N=53) | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 (N=55) | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 (N=56) | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 (N=55) | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 (N=37) | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 (N=56) | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 (N=54) | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 (N=38) | Part 1 Cohort B7: mRNA-1083.3 (N=54) | Part 2: Influenza Vaccine 1 (N=40) | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 (N=39) | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 (N=40) | Part 2: COVID-19 Vaccine 2 (N=42) | Part 2: Investigational COVID-19 Vaccine 2 (N=40) | Part 2: mRNA-1083 Composition 1 Dose Level 1 (N=40) | Part 2: mRNA-1083 Composition 1 Dose Level 2 (N=42) | Part 2: mRNA-1083 Composition 1 Dose Level 3 (N=41) | Part 2: mRNA-1083 Composition 1 Dose Level 4 (N=41) | Part 2: mRNA-1083 Composition 2 Dose Level 1 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 2 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 3 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 4 (N=42)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar II disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pseudoaneurysm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Of all the SAEs reported in this study, only the SAE of Hepatic Enzyme Increased in the Influenza Vaccine 2 group was considered related to the study injection by the Investigator.
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort A12: Influenza Vaccine 1 (N=54) | Part 1 Cohort A13: Influenza Vaccine 2 (N=53) | Part 1 Cohort A11: Investigational Influenza Vaccine 2 (N=54) | Part 1 Cohort A8: Investigational Influenza Vaccine 1 (N=51) | Part 1 Cohort A10: COVID-19 Vaccine 1 (N=54) | Part 1 Cohort A9: Investigational COVID-19 Vaccine 1 (N=52) | Part 1 Cohort A2: mRNA-1083.1 Dose Level 2 (N=51) | Part 1 Cohort A3: mRNA-1083.1 Dose Level 3 (N=33) | Part 1 Cohort A4: mRNA-1083.2 Dose Level 1 (N=55) | Part 1 Cohort A5: mRNA-1083.2 Dose Level 2 (N=53) | Part 1 Cohort A6: mRNA-1083.2 Dose Level 3 (N=33) | Part 1 Cohort A7: mRNA-1083.3 (N=53) | Part 1 Cohort B12: Influenza Vaccine 1 (N=52) | Part 1 Cohort B11: Investigational Influenza Vaccine 2 (N=55) | Part 1 Cohort B8: Investigational Influenza Vaccine 1 (N=55) | Part 1 Cohort B10: COVID-19 Vaccine 1 (N=53) | Part 1 Cohort B9: Investigational COVID-19 Vaccine 1 (N=55) | Part 1 Cohort B1: mRNA-1083.1 Dose Level 1 (N=56) | Part 1 Cohort B2: mRNA-1083.1 Dose Level 2 (N=55) | Part 1 Cohort B3: mRNA-1083.1 Dose Level 3 (N=37) | Part 1 Cohort B4: mRNA-1083.2 Dose Level 1 (N=56) | Part 1 Cohort B5: mRNA-1083.2 Dose Level 2 (N=54) | Part 1 Cohort B6: mRNA-1083.2 Dose Level 3 (N=38) | Part 1 Cohort B7: mRNA-1083.3 (N=54) | Part 2: Influenza Vaccine 1 (N=40) | Part 2: Investigational Influenza Vaccine 1 Dose Level 1 (N=39) | Part 2: Investigational Influenza Vaccine 1 Dose Level 2 (N=40) | Part 2: COVID-19 Vaccine 2 (N=42) | Part 2: Investigational COVID-19 Vaccine 2 (N=40) | Part 2: mRNA-1083 Composition 1 Dose Level 1 (N=40) | Part 2: mRNA-1083 Composition 1 Dose Level 2 (N=42) | Part 2: mRNA-1083 Composition 1 Dose Level 3 (N=41) | Part 2: mRNA-1083 Composition 1 Dose Level 4 (N=41) | Part 2: mRNA-1083 Composition 2 Dose Level 1 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 2 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 3 (N=40) | Part 2: mRNA-1083 Composition 2 Dose Level 4 (N=42)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 6 (8) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT05827926/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT05827926/SAP_001.pdf